CLINICAL TRIAL: NCT00839254
Title: Impact on Nasopharyngeal Carriage, Acute Otitis Media, Immunogenicity and Safety of GSK Biologicals' Pneumococcal Conjugate Vaccine 1024850A
Brief Title: Impact on Carriage, Acute Otitis Media, Immuno & Safety of GSK Biologicals' Pneumococcal Conjugate Vaccine 1024850A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112595; 2008-006551-51 (EudraCT Number)
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae
Keywords: Streptococcus pneumoniae; acute otitis media; Pneumococcal conjugate vaccine; nasopharyngeal carriage; Haemophilus influenzae; immunogenicity; invasive disease
MeSH Terms: conditions — Streptococcal Infections; Otitis Media; Haemophilus Infections | interventions — Hepatitis B Vaccines; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- 10Pn3+1-6W-6M/053 Group (Experimental): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
  Interventions: Biological: Pneumococcal conjugate vaccine Synflorix (GSK1024850A)
- 10Pn2+1-6W-6M/053 Group (Experimental): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
  Interventions: Biological: Pneumococcal conjugate vaccine Synflorix (GSK1024850A)
- Ctrl3+1-6W-6M/053 Group (Active Comparator): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B vaccine (called also HBV vaccine) according to a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
  Interventions: Biological: GSK Biologicals' Engerix TM vaccine (Hepatitis B vaccine)
- Ctrl2+1-6W-6M/053 Group (Active Comparator): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B vaccine (called also HBV vaccine) according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
  Interventions: Biological: GSK Biologicals' Engerix TM vaccine (Hepatitis B vaccine)
- 10Pn7-11M/053 Group (Experimental): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 7 to 11 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (7-11M Schedule). The vaccine was administered intramuscularly in the thigh or in the deltoid region of upper arm, provided the muscle size was adequate.
  Interventions: Biological: Pneumococcal conjugate vaccine Synflorix (GSK1024850A)
- Ctrl7-11M/053 Group (Active Comparator): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 7 to 11 months at enrolment. Subjects received the Engerix B (called also HBV) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (7-11M Schedule). The vaccine was administered intramuscularly in the thigh or in the deltoid region of upper arm, provided the muscle size was adequate.
  Interventions: Biological: GSK Biologicals' Engerix TM vaccine (Hepatitis B vaccine)
- 10Pn12-18M/053 Group (Active Comparator): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 12 to 18 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). The vaccine was administered intramuscularly in the thigh or in the deltoid region of upper arm, provided the muscle size was adequate.
  Interventions: Biological: Pneumococcal conjugate vaccine Synflorix (GSK1024850A)
- Ctrl12-18M/053 Group (Experimental): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 12 to 18 months at enrolment. Subjects received the Havrix (called also HAV) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). The vaccine was administered intramuscularly in the thigh or in the deltoid region of upper arm, provided the muscle size was adequate.
  Interventions: Biological: GSK Biologicals' Havrix TM vaccine (Hepatitis A vaccine)

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine Synflorix (GSK1024850A) — 2, 3 or 4 Intramuscular injections, depending on the age at the time of first vaccination
  Arms: 10Pn12-18M/053 Group; 10Pn2+1-6W-6M/053 Group; 10Pn3+1-6W-6M/053 Group; 10Pn7-11M/053 Group
Biological: GSK Biologicals' Engerix TM vaccine (Hepatitis B vaccine) — 3 or 4 Intramuscular injections, depending on the age at the time of first vaccination only for children < 12 months of age at the time of first study vaccination.
  Arms: Ctrl2+1-6W-6M/053 Group; Ctrl3+1-6W-6M/053 Group; Ctrl7-11M/053 Group
Biological: GSK Biologicals' Havrix TM vaccine (Hepatitis A vaccine) — 2 Intramuscular injections only for children >= 12 months of age at the time of first study vaccination.
  Arms: Ctrl12-18M/053 Group

SUMMARY:
The aim of this study is to assess the effectiveness of GSK Biologicals' pneumococcal conjugate vaccine (GSK1024850A) in preventing invasive disease caused by S. pneumoniae or H. influenzae and in reducing occurrence of hospital-diagnosed pneumonia cases, tympanostomy tube placement and outpatient antimicrobial prescriptions in children starting vaccination below 18 months of age. These data will be collected from the national registers and will be analyzed in combination with data collected for subjects enrolled in a large scale cluster-randomized study 111442.

The study will also assess the immune response to the GSK1024850A vaccine and the impact of the vaccine on occurrence of acute otitis media, carriage, safety in children starting vaccination below 18 months of age.

DETAILED DESCRIPTION:
The protocol posting has been updated with regards to the outcome measures following Protocol amendment 4, 12 August 2011.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol should be enrolled in the study.
* Male or female between, and including, 6 weeks to 18 months of age at the time of the first vaccination.
* Written informed consent obtained from parent(s) or from the guardian(s) of the subject.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first dose of study vaccine, or planned use of such a vaccine(s) other than the study vaccine(s) during the entire study period.
* Previous vaccination with any registered, non-registered or investigational pneumococcal vaccine, or planned use of such a vaccine other than the study vaccine during the study period. If a child belongs to a high risk group for pneumococcal infections (such as children with an anatomic or functional asplenia, HIV infection, chronic cardiac or respiratory disease (not asthma), diabetes, cochlear implant, CSF fistula or with significant immunodeficiency) for which a licensed pneumococcal conjugate vaccine is made locally available, the subject can not be enrolled in the study and should be referred to the specific immunization program.
* Previous vaccination against Hepatitis B virus with any registered, non-registered or investigational vaccine, or planned use of such a vaccine other than the study vaccine during the study period.
* Previous vaccination against Hepatitis A virus with any registered, non-registered or investigational vaccine, or planned use of such a vaccine other than the study vaccine during the study period.
* Known severe hypersensitivity to any component of the study vaccines, including neomycin.
* Any medical condition that would contraindicate the initiation of routine immunization outside a clinical trial context.

Ages: 6 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6181 (Actual)
Dates: Start 2009-02-18 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2012-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Finland (13):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=4324

REFERENCES:
- [Background] Vesikari T, Forsten A, Seppa I, Kaijalainen T, Puumalainen T, Soininen A, Traskine M, Lommel P, Schoonbroodt S, Hezareh M, Moreira M, Borys D, Schuerman L. Effectiveness of the 10-Valent Pneumococcal Nontypeable Haemophilus influenzae Protein D-Conjugated Vaccine (PHiD-CV) Against Carriage and Acute Otitis Media-A Double-Blind Randomized Clinical Trial in Finland. J Pediatric Infect Dis Soc. 2016 Sep;5(3):237-248. doi: 10.1093/jpids/piw010. Epub 2016 Apr 28. PMID 27125273
- [Derived] Rinta-Kokko H, Palmu AA, Ruokokoski E, Nieminen H, Moreira M, Schuerman L, Borys D, Jokinen J. Evaluation of the indirect impact of the 10-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine in a cluster-randomised trial. PLoS One. 2022 Jan 5;17(1):e0261750. doi: 10.1371/journal.pone.0261750. eCollection 2022. PMID 34986178
- [Derived] Nieminen H, Rinta-Kokko H, Jokinen J, Puumalainen T, Moreira M, Borys D, Schuerman L, Palmu AA. Effectiveness of the 10-valent pneumococcal conjugate vaccine among girls, boys, preterm and low-birth-weight infants - Results from a randomized, double-blind vaccine trial. Vaccine. 2019 Jun 19;37(28):3715-3721. doi: 10.1016/j.vaccine.2019.05.033. Epub 2019 May 20. PMID 31122856
- [Derived] Kilpi TM, Jokinen J, Puumalainen T, Nieminen H, Ruokokoski E, Rinta-Kokko H, Traskine M, Lommel P, Moreira M, Ruiz-Guinazu J, Borys D, Schuerman L, Palmu AA. Effectiveness of pneumococcal Haemophilus influenzae protein D conjugate vaccine against pneumonia in children: A cluster-randomised trial. Vaccine. 2018 Sep 18;36(39):5891-5901. doi: 10.1016/j.vaccine.2018.08.020. Epub 2018 Aug 23. PMID 30145098
- [Derived] Palmu AA, Jokinen J, Nieminen H, Rinta-Kokko H, Ruokokoski E, Puumalainen T, Moreira M, Schuerman L, Borys D, Kilpi TM. Vaccine-preventable disease incidence of pneumococcal conjugate vaccine in the Finnish invasive pneumococcal disease vaccine trial. Vaccine. 2018 Mar 27;36(14):1816-1822. doi: 10.1016/j.vaccine.2018.02.088. PMID 29503110
- [Derived] Palmu AA, Jokinen J, Nieminen H, Rinta-Kokko H, Ruokokoski E, Puumalainen T, Traskine M, Moreira M, Borys D, Schuerman L, Kilpi TM. Effectiveness of the Ten-valent Pneumococcal Conjugate Vaccine Against Tympanostomy Tube Placements in a Cluster-randomized Trial. Pediatr Infect Dis J. 2015 Nov;34(11):1230-5. doi: 10.1097/INF.0000000000000857. PMID 26284652
- [Derived] Palmu AA, Jokinen J, Nieminen H, Syrjanen R, Ruokokoski E, Puumalainen T, Moreira M, Schuerman L, Borys D, Kilpi TM. Vaccine effectiveness of the pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10) against clinically suspected invasive pneumococcal disease: a cluster-randomised trial. Lancet Respir Med. 2014 Sep;2(9):717-27. doi: 10.1016/S2213-2600(14)70139-0. Epub 2014 Aug 7. PMID 25127244
- [Derived] Palmu AA, Jokinen J, Nieminen H, Rinta-Kokko H, Ruokokoski E, Puumalainen T, Borys D, Lommel P, Traskine M, Moreira M, Schuerman L, Kilpi TM. Effect of pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10) on outpatient antimicrobial purchases: a double-blind, cluster randomised phase 3-4 trial. Lancet Infect Dis. 2014 Mar;14(3):205-12. doi: 10.1016/S1473-3099(13)70338-4. Epub 2013 Nov 26. PMID 24287186
- [Derived] Palmu AA, Jokinen J, Borys D, Nieminen H, Ruokokoski E, Siira L, Puumalainen T, Lommel P, Hezareh M, Moreira M, Schuerman L, Kilpi TM. Effectiveness of the ten-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10) against invasive pneumococcal disease: a cluster randomised trial. Lancet. 2013 Jan 19;381(9862):214-22. doi: 10.1016/S0140-6736(12)61854-6. Epub 2012 Nov 16. PMID 23158882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is linked with 10PN-PD-DIT-043 (111442) study (NCT00861380.-EudraCT: 2008-005149-48) with which primary objectives and outcomes are common. Subjects of 10PN-PD-DIT-043 study contributed to the results of this study.
Pre-assignment Details: Out of 6183 subjects enrolled, 6177 were analyzed:(6174 subjects and 3 of them received 2 subject numbers, without any impact on the results of the analyses. Total population assessed for combined analyses performed on both studies included 45977 subjects, see details in groups description.
Groups:
- Ctrl3+1-6W-6M/053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B (called also HBV vaccine) according to a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
- Ctrl2+1-6W-6M/053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) study, aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B (called also HBV vaccine) according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
Period: Overall Study
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Started | 1849 | 1316 | 1069 | 859 | 241 | 204 | 368 | 271
Completed | 1696 | 1224 | 979 | 797 | 204 | 178 | 340 | 256
Not Completed | 153 | 92 | 90 | 62 | 37 | 26 | 28 | 15
Not completed — Protocol Violation | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Wrong treatment number allocation | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 12 | 6 | 3 | 5 | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 87 | 53 | 54 | 32 | 27 | 15 | 22 | 9
Not completed — Wrong group allocation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Parents wanted pneumococcal vaccine | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawn due to non-compliance | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 51 | 30 | 32 | 24 | 8 | 8 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group | Total
Number analyzed (Participants) | 1849 | 1316 | 1069 | 859 | 241 | 204 | 368 | 271 | 6177
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.4 (1.02) | 2.3 (0.95) | 2.6 (1.19) | 2.4 (1) | 9 (1.44) | 8.7 (1.39) | 15 (1.99) | 15.2 (1.99) | 7.2 (1.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 921 | 681 | 551 | 393 | 118 | 113 | 173 | 142 | 3092
  Male | 928 | 635 | 518 | 466 | 123 | 91 | 195 | 129 | 3085
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage / African American | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 5
  White - Arabic / north African heritage | 7 | 5 | 4 | 6 | 3 | 0 | 2 | 0 | 27
  White - Caucasian / European heritage | 1822 | 1303 | 1058 | 845 | 235 | 201 | 362 | 270 | 6096
  Unspecified | 19 | 8 | 7 | 8 | 2 | 2 | 2 | 1 | 49

OUTCOME MEASURES:

1. Primary Outcome: Person Year Rate as Regards Subjects With Culture-confirmed IPD Due to Any of the 10 Pneumococcal Vaccine Serotypes. In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course.
Description: The PYAR (Person-Year Rate) as regards subjects with culture-confirmed invasive pneumococcal disease (IPD) due to any of the pneumococcal vaccine serotypes was tabulated (vaccine pneumococcal serotypes = serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F). PYAR was calculated as follows n (= number of subjects reported with a culture confirmed IPD) divided by T (= sum of follow-up period expressed in years) (per 1000) as well as the corresponding 95% confidence interval (CI), calculated as a 2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata.
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end of the blinded invasive disease (ID) Follow-up period (The blinded ID Follow-up period lasted at least 30 months).
Population: The analysis was performed on the Infant Vaccinated cohort, including all vaccinated, subjects in the 10PN-PD-DIT-043 NCT00839254 study and vaccinated subjects of 10PN-PD-DIT-053 NCT00839254 study contributing to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 3-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn3+1-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 8427 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule). Refer to group description for 10Pn3+1-6W-6M/053 Group for details on vaccine specifics and administration route in this group.
- Ctrl-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 8872 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B (called also HBV vaccine) according to either a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule), or according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group descriptions for Ctrl3+1-6W-6M/053 and Ctrl2+1-6W-6M/053 groups for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10201
Participants per 1000 person-years | 0.000 [0.000 to 0.172] | 0.564 [0.291 to 0.984]
Statistical Analysis 1: Comparison: 10Pn3+1-6W-6M/043+053 Group vs Ctrl-6W-6M/043+053 Group; Analysis aimed at providing an estimate of vaccine effectiveness (VE) at preventing culture-confirmed IPD by comparing PYARs between groups taking into account the following parameters: T, n, n+ (number of clusters with at least one event culture-confirmed ID), and n/T. VE of the 10Pn vaccine in preventing culture-confirmed IPD due to the 10 vaccine serotypes was demonstrated if the 2-sided p-value calculated for the null hypothesis H0 = (vaccine-type [VT] IPD VE = 0%) was lower than (<) 5%; Test type: Superiority — VE (defined as 1 minus Relative Risk (RR)) was calculated by comparing numbers of culture-confirmed IPD. The number of subjects with IPD in each cluster was compared between groups (10PN3+1 vs Control). This comparison was done using a negative binomial log-linear model with correction for dispersion group- and cluster-related effect; p < 0.0001, Regression, Linear — P-value was calculated using a classical log linear Poisson regression with strata, without taking into account the multiplicity of the endpoints; VE (1-RR) = 100, 95% CI 2-sided [82.8 to 100]

2. Primary Outcome: Person Year Rate as Regards Subjects With Culture-confirmed IPD Due to Any of the 10 Pneumococcal Vaccine Serotypes. In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 2-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn2+1-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 9112 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group description for 10Pn2+1-6W-6M/053 Group for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10201
Participants per 1000 person-years | 0.048 [0.001 to 0.270] | 0.564 [0.291 to 0.984]
Statistical Analysis 1: Comparison: 10Pn2+1-6W-6M/043+053 Group vs Ctrl-6W-6M/043+053 Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — VE (defined as 1 minus Relative Risk (RR)) was calculated by comparing numbers of culture-confirmed IPD. The number of subjects with IPD in each cluster was compared between groups (10PN2+1 vs Control). This comparison was done using a negative binomial log-linear model with correction for dispersion group- and cluster-related effect; p = 0.0009, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; VE (1-RR) = 91.8, 95% CI 2-sided [58.3 to 99.6]

3. Secondary Outcome: Person Year Rate in the Prevention of Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course.
Description: The PYAR (Person-Year Rate) was calculated as follows n (= number of subjects reported with a culture confirmed IPD) divided by T (= sum of follow-up period expressed in years) (per 1000) as well as the corresponding 95% confidence interval (CI), calculated as a 2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata.
Time Frame: as for outcome 1
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 3-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10201
Participants per 1000 person-years
  Culture confirmed ID | 0.093 [0.011 to 0.336] | 0.845 [0.501 to 1.336]
  Pneumococcal invasive disease (IPD) | 0.000 [0.000 to 0.172] | 0.657 [0.359 to 1.103]
  Serotype 4 | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  Serotype 6B | 0.000 [0.000 to 0.172] | 0.235 [0.076 to 0.548]
  Serotype 7F | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  Serotype 14 | 0.000 [0.000 to 0.172] | 0.188 [0.051 to 0.481]
  Serotype 18C | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Serotype 19F | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Serotype 23F | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Cross-reactive serotypes | 0.000 [0.000 to 0.172] | 0.094 [0.011 to 0.339]
  Serotype 6A | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Serotype 19A | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Other pneumococcal serotypes | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  Serotype 3 | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  Serotype 15C | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  H. influenzae ID | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Non-typeable (NTHI) | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Other bacteria | 0.093 [0.011 to 0.336] | 0.188 [0.051 to 0.481]
  Neisseria meningitidis | 0.093 [0.011 to 0.336] | 0.047 [0.001 to 0.262]
  Streptococcus pyogenes | 0.000 [0.000 to 0.172] | 0.094 [0.011 to 0.339]
  Moraxella catarrhalis | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]

4. Secondary Outcome: Person Year Rate in the Prevention of Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course.
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10201
Participants per 1000 person-years
  Culture confirmed ID | 0.194 [0.053 to 0.496] | 0.845 [0.501 to 1.336]
  Pneumococcal invasive disease (IPD) | 0.097 [0.012 to 0.350] | 0.657 [0.359 to 1.103]
  Vaccine serotypes (vaccine type-IPD) | 0.048 [0.001 to 0.270] | 0.564 [0.291 to 0.984]
  Serotype 4 | 0.000 [0.000 to 0.179] | 0.000 [0.000 to 0.173]
  Serotype 6B | 0.000 [0.000 to 0.179] | 0.235 [0.076 to 0.548]
  Serotype 7F | 0.048 [0.001 to 0.270] | 0.000 [0.000 to 0.173]
  Serotype 14 | 0.000 [0.000 to 0.179] | 0.188 [0.051 to 0.481]
  Serotype 18C | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Serotype 19F | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Serotype 23F | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Cross-reactive serotypes | 0.000 [0.000 to 0.179] | 0.094 [0.011 to 0.339]
  Serotype 6A | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Serotype 19A | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Other pneumococcal serotypes | 0.048 [0.001 to 0.270] | 0.000 [0.000 to 0.173]
  Serotype 3 | 0.048 [0.001 to 0.270] | 0.000 [0.000 to 0.173]
  Serotype 15C | 0.000 [0.000 to 0.179] | 0.000 [0.000 to 0.173]
  H. influenzae ID | 0.048 [0.001 to 0.270] | 0.047 [0.001 to 0.262]
  Non-typeable (NTHI) | 0.048 [0.001 to 0.270] | 0.047 [0.001 to 0.262]
  Other bacteria | 0.048 [0.001 to 0.270] | 0.188 [0.051 to 0.481]
  Neisseria meningitidis | 0.048 [0.001 to 0.270] | 0.047 [0.001 to 0.262]
  Streptococcus pyogenes | 0.000 [0.000 to 0.179] | 0.094 [0.011 to 0.339]
  Moraxella catarrhalis | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]

5. Secondary Outcome: Person Year Rate in the Prevention of Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination in the 7-11 Months Schedule.
Description: as for outcome 3
Time Frame: as for outcome 1
Population: The analysis was performed on the Catch-up Vaccinated cohort, which included all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with a 2-dose primary vaccination between 7 and 11 months of age.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 3689 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 7 to 11 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (7-11M Schedule). Refer to group description for 10Pn7-11M/053 Group for details on vaccine specifics and administration route in this group.
- Ctrl7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 1812 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 7 to 11 months at enrolment. Subjects received the Engerix B (called also HBV) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (7-11M Schedule). Refer to group description for Ctrl7-11M/053 Group for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1908
Participants per 1000 person-years
  Culture confirmed ID | 0.000 [0.000 to 0.410] | 0.446 [0.054 to 1.612]
  Pneumococcal invasive disease (IPD) | 0.000 [0.000 to 0.410] | 0.446 [0.054 to 1.612]
  Vaccine serotypes (vaccine type-IPD) | 0.000 [0.000 to 0.410] | 0.446 [0.054 to 1.612]
  Serotype 4 | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 6B | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 7F | 0.000 [0.000 to 0.410] | 0.223 [0.006 to 1.243]
  Serotype 14 | 0.000 [0.000 to 0.410] | 0.223 [0.006 to 1.243]
  Serotype 18C | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 19F | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 23F | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Cross-reactive serotypes | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 6A | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 19A | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Other pneumococcal serotypes | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 3 | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 15C | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  H. influenzae ID | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Non-typeable (NTHI) | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Other bacteria | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]

6. Secondary Outcome: Person Year Rate in the Prevention of Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination in the 12-18 Months Schedule.
Description: as for outcome 3
Time Frame: as for outcome 1
Population: The analysis was performed on the Catch-up Vaccinated cohort, which included all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with a 2-dose primary vaccination between 12 and 18 months of age.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn12-18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 6249 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 12 to 18 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for 10Pn12-18M/053 Group for details on vaccine specifics and administration route in this group.
- Ctrl12-18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 3020 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 12 to 18 months at enrolment. Subjects received the Havrix (called also HAV) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for Ctrl12-18M/053 Group for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6535 | 3126
Participants per 1000 person-years
  Culture confirmed ID | 0.000 [0.000 to 0.240] | 0.674 [0.219 to 1.572]
  Pneumococcal invasive disease (IPD) | 0.000 [0.000 to 0.240] | 0.674 [0.219 to 1.572]
  Vaccine serotypes (vaccine type-IPD) | 0.000 [0.000 to 0.240] | 0.404 [0.083 to 1.181]
  Serotype 4 | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  Serotype 6B | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  Serotype 7F | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 14 | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 18C | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 19F | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  Serotype 23F | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Cross-reactive serotypes | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 6A | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 19A | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Other pneumococcal serotypes | 0.000 [0.000 to 0.240] | 0.269 [0.033 to 0.974]
  Serotype 3 | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  Serotype 15C | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  H. influenzae ID | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Non-typeable (NTHI) | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Other bacteria | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]

7. Secondary Outcome: Person Year Rate in the Prevention of Probable Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course.
Description: The PYAR (Person-Year Rate) was calculated as follows n (= number of subjects reported with a probable or culture confirmed ID) divided by T (= sum of follow-up period expressed in years) (per 1000) as well as the corresponding 95% confidence interval (CI), calculated as a 2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata.
Time Frame: as for outcome 1
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 3-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10201
Participants per 1000 person-years
  Probable cases of IPD | 0.000 [0.000 to 0.172] | 0.141 [0.029 to 0.412]
  Confirmed or probable cases of IPD | 0.000 [0.000 to 0.172] | 0.798 [0.465 to 1.278]

8. Secondary Outcome: Person Year Rate in the Prevention of Probable or Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course.
Description: as for outcome 7
Time Frame: as for outcome 1
Population: The analysis was performed on the Infant Vaccinated cohort, all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 2-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- Ctrl-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 8872 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B vaccine (called also HBV vaccine) according to either a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule), or according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group descriptions for Ctrl3+1-6W-6M/053 and Ctrl2+1-6W-6M/053 groups for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10201
Participants per 1000 person-years
  Probable cases of IPD | 0.000 [0.000 to 0.179] | 0.141 [0.029 to 0.412]
  Confirmed or probable cases of IPD | 0.097 [0.012 to 0.350] | 0.798 [0.465 to 1.278]

9. Secondary Outcome: Person Year Rate in the Prevention of Probable or Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination in the 7-11 Months Schedule.
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1908
Participants per 1000 person-years
  Probable cases of IPD | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Confirmed or probable cases of IPD | 0.000 [0.000 to 0.410] | 0.446 [0.054 to 1.612]

10. Secondary Outcome: Person Year Rate in the Prevention of Probable or Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination in the 12-18 Months Schedule.
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6535 | 3126
Participants per 1000 person-years
  Probable cases of IPD | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Confirmed or probable cases of IPD | 0.000 [0.000 to 0.240] | 0.674 [0.219 to 1.572]

11. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course.
Description: PYAR was calculated: n (= number of subjects with hospital-diagnosed pneumonia) divided by T (= sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. Hospital-diagnosed pneumonia (HDP) cases identified based on hospital discharge diagnosis using international Classification of Disease (ICD)-10 diagnosis codes: J10.0 (Influenza with HDP, other influenza virus identified), J11.0 (Influenza with HDP, virus not identified), J12 (Viral HDP, not elsewhere classified), J13 (HDP due to Sp.), J14 (for HDP due to Hi.), J15 (all HDP, not elsewhere classified), J16 (HDP due to other infectious organisms, not elsewhere classified), J17 (HDP in diseases classified elsewhere), J18 (HDP organism unspecified), J85.1 (Abscess of lung with HDP), and J86 (Pyothorax including empyema).
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end date of the follow-up (31 December 2011) - FU mean time=24 months.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10200
Participants per 1000 person-years | 10.131 [8.804 to 11.601] | 13.854 [12.287 to 15.566]

12. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course.
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10200
Participants per 1000 person-years | 10.155 [8.800 to 11.660] | 13.854 [12.287 to 15.566]

13. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia- In Children Starting Vaccination in the 7-11 Months Schedule.
Description: as for outcome 11
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end date of the follow-up (31 December 2011) - FU mean time=27 months.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1907
Participants per 1000 person-years | 10.263 [8.242 to 12.630] | 15.752 [12.232 to 19.970]

14. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia - In Children Starting Vaccination in the 12-18 Months Schedule.
Description: as for outcome 11
Time Frame: as for outcome 13
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6534 | 3126
Participants per 1000 person-years | 9.322 [7.832 to 11.013] | 11.739 [9.363 to 14.533]

15. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia With Chest X-ray (CXR) Reading According to WHO Criteria- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course.
Description: PYAR was calculated: n (= number of subjects with hospital-diagnosed pneumonia [HDP]) divided by T (= sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata for non-consolidated HDP and without strata for consolidated HDP). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. CXR HDP was defined as a HDP case with the presence of abnormal pulmonary infiltrates on the CXR as per independent review panel judgement using WHO methodology. Abnormal pulmonary infiltrates could be either with (Consolidated HDP) or without (Non-consolidated HDP) alveolar consolidation/pleural effusion. New cases of HDP and CXR HDP were based on a 30-day rule, i.e. a new episode was considered if at least a 30-day interval elapsed from the onset of the previous episode.
Time Frame: as for outcome 11
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10200
Participants per 1000 person-years
  Consolidated pneumonia | 2.181 [1.591 to 2.919] | 3.965 [3.149 to 4.929]
  Non-consolidated pneumonia | 2.908 [2.219 to 3.744] | 2.937 [2.241 to 3.781]
  Consolidated or non-consolidated pneumonia | 5.090 [4.163 to 6.161] | 6.903 [5.810 to 8.141]

16. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia With CXR Reading According to WHO Criteria - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course.
Description: as for outcome 15
Time Frame: as for outcome 11
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 2-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10200
Participants per 1000 person-years
  Consolidated pneumonia | 2.273 [1.658 to 3.042] | 3.965 [3.149 to 4.929]
  Non-consolidated pneumonia | 2.627 [1.962 to 3.445] | 2.937 [2.241 to 3.781]
  Consolidated or non-consolidated pneumonia | 4.901 [3.974 to 5.978] | 6.903 [5.810 to 8.141]

17. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia With CXR Reading According to WHO Criteria - In Children Starting Vaccination in the 7-11 Months Schedule.
Description: as for outcome 15
Time Frame: as for outcome 13
Population: The analysis was performed on the Catch-up Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with a 2-dose primary vaccination between 7 and 11 months of age.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 3689 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 7 to 11 months at enrolment. Subjects received the Synflorix (called aslo 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (7-11M Schedule). Refer to group description for 10Pn7-11M/053 Group for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1907
Participants per 1000 person-years
  Consolidated pneumonia | 1.960 [1.142 to 3.139] | 4.401 [2.650 to 6.873]
  Non-consolidated pneumonia | 3.344 [2.240 to 4.803] | 4.865 [3.011 to 7.436]
  Consolidated or non-consolidated pneumonia | 5.305 [3.884 to 7.076] | 9.266 [6.620 to 12.618]

18. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia With CXR Reading According to WHO Criteria - In Children Starting Vaccination in the 12-18 Months Schedule.
Description: as for outcome 15
Time Frame: as for outcome 13
Population: The analysis was performed on the Catch-up Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with a 2-dose primary vaccination between 12 and 18 months of age.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6534 | 3126
Participants per 1000 person-years
  Consolidated pneumonia | 1.824 [1.202 to 2.654] | 3.494 [2.261 to 5.157]
  Non-consolidated pneumonia | 2.837 [2.045 to 3.835] | 2.935 [1.817 to 4.486]
  Consolidated or non-consolidated pneumonia | 4.661 [3.626 to 5.899] | 6.428 [4.706 to 8.574]

19. Secondary Outcome: Person Year Rate in Prevention of All Tympanostomy Tube Placements- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course.
Description: PYAR was calculated: n (= number of subjects with tympanostomy tube placement[TTP]) divided by T (= sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. A TTP episode was defined as a TTP episode classified under the DCA 20 code in the Finnish National Institute of Health and Welfare (THL) and Social Insurance Institution of Finland (KELA) registers, using the Nordic Centre for Classifications in Health Care (NOMESCO) Classification of Surgical Procedures (NCSP), version 1.12 from January 2008, and could refer to either an unilateral or a bilateral TTP procedure. New episodes of TTP defined according to a 30-day rule meaning that a new episode was considered if at least 30-day interval elapsed from the onset of the previous episode.
Time Frame: as for outcome 11
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10200
Participants per 1000 person-years | 68.735 [65.203 to 72.408] | 79.504 [75.683 to 83.467]

20. Secondary Outcome: Person Year Rate in Prevention of All Tympanostomy Tube Placements - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course.
Description: as for outcome 19
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10200
Participants per 1000 person-years | 66.083 [62.550 to 69.764] | 79.504 [75.683 to 83.467]

21. Secondary Outcome: Person Year Rate in Prevention of All Tympanostomy Tube Placements - In Children Starting Vaccination in the 7-11 Months Schedule.
Description: as for outcome 19
Time Frame: as for outcome 13
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1907
Participants per 1000 person-years | 68.153 [62.769 to 73.876] | 79.920 [71.708 to 88.814]

22. Secondary Outcome: Person Year Rate in Prevention of All Tympanostomy Tube Placements - In Children Starting Vaccination in the 12-18 Months Schedule.
Description: as for outcome 19
Time Frame: as for outcome 13
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6534 | 3126
Participants per 1000 person-years | 56.809 [53.034 to 60.782] | 58.973 [53.480 to 64.877]

23. Secondary Outcome: Person Year Rate in Prevention of All Antimicrobial Prescriptions- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course.
Description: PYAR was calculated: n (= number of subjects with antimicrobial prescriptions (APs)) divided by T (= sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. An APs episode was an episode of APs to an infant/child falling under following Anatomic Therapeutic Chemical [ATC] codes: J01 (APs) and following codes for AP usually recommended for otitis media (OM) and respiratory tract infections (RTI). "For OM and RTI" category corresponds to following definition: APs for antibacterial usually recommended for OM and RTI (ATC codes: J01CA04, J01CR02, J01CE02, J01DC02, J01DC04, J01EE02, J01FA09 and J01FA10). New episodes of APs were analyzed according to a 2-day rule meaning new episode considered if at least 2 day interval elapsed from the onset of the previous episode.
Time Frame: as for outcome 11
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10200
Participants per 1000 person-years
  Antimicrobial prescriptions (ATC code J01) | 1592.585 [1575.411 to 1609.901] | 1706.194 [1688.328 to 1724.202]
  For otitis media and respiratory infections | 1451.141 [1434.749 to 1467.674] | 1565.692 [1548.579 to 1582.947]

24. Secondary Outcome: Person Year Rate in Prevention of All Antimicrobial Prescriptions - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course.
Description: as for outcome 23
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10200
Participants per 1000 person-years
  Antimicrobial prescriptions (ATC code J01) | 1552.493 [1535.183 to 1569.950] | 1706.194 [1688.328 to 1724.202]
  For otitis media and respiratory infections | 1415.983 [1399.453 to 1432.659] | 1565.692 [1548.579 to 1582.947]

25. Secondary Outcome: Person Year Rate in Prevention of All Antimicrobial Prescriptions - In Children Starting Vaccination in the 7-11 Months Schedule.
Description: as for outcome 23
Time Frame: as for outcome 13
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1907
Participants per 1000 person-years
  Antimicrobial prescriptions (ATC code J01) | 1536.618 [1510.637 to 1562.934] | 1649.360 [1611.269 to 1688.124]
  For otitis media and respiratory infections | 1390.856 [1366.143 to 1415.903] | 1499.713 [1463.401 to 1536.698]

26. Secondary Outcome: Person Year Rate in Prevention of All Antimicrobial Prescriptions - In Children Starting Vaccination in the 12-18 Months Schedule.
Description: as for outcome 23
Time Frame: as for outcome 13
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6534 | 3126
Participants per 1000 person-years
  Antimicrobial prescriptions (ATC code J01) | 1315.936 [1297.521 to 1334.547] | 1421.774 [1394.280 to 1449.675]
  For otitis media and respiratory infections | 1177.729 [1160.312 to 1195.343] | 1271.268 [1245.277 to 1297.665]

27. Secondary Outcome: Number of Subjects Classified by Antimicrobial Susceptiblity of IPD Isolates in Children Starting Vaccination Within 7 Months of Life and Assigned to a 2 or 3-dose Primary Vaccination Course
Description: Antimicrobial susceptibility classification of IPD isolates reported during IPD follow-up with percentages for each serotype for the following categories: S= susceptible; I = intermediate ; R = resistant; N = not available.
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end date of the follow-up (31 December 2011) - mean FU time=24 months.
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 0 | 2 | 24
Participants
  Serotype-4 -Pencillin-S |  | 0 | 1
  Serotype-6A -Pencillin-S |  | 0 | 1
  Serotype-6B -Pencillin-I |  | 0 | 3
  Serotype-6B -Pencillin-R |  | 0 | 1
  Serotype-6B -Pencillin-S |  | 0 | 2
  Serotype-7F -Pencillin-S |  | 1 | 1
  Serotype-14 -Pencillin-I |  | 0 | 2
  Serotype-14 -Pencillin-R |  | 0 | 1
  Serotype-14 -Pencillin-S |  | 0 | 2
  Serotype-15C -Pencillin-S |  | 0 | 1
  Serotype-18C -Pencillin-S |  | 0 | 1
  Serotype-19A -Pencillin-I |  | 0 | 1
  Serotype-19F -Pencillin-I |  | 0 | 1
  Serotype-19F -Pencillin-S |  | 0 | 1
  Serotype-23F -Pencillin-S |  | 0 | 1
  Serotype-N -Pencillin-N |  | 1 | 4
  Serotype-4 -Erythromycin-S |  | 0 | 1
  Serotype-6A -Erythromycin-S |  | 0 | 1
  Serotype-6B -Erythromycin-R |  | 0 | 5
  Serotype-6B -Erythromycin-S |  | 0 | 1
  Serotype-7F -Erythromycin-S |  | 1 | 1
  Serotype-14 -Erythromycin-R |  | 0 | 4
  Serotype-14 -Erythromycin-S |  | 0 | 1
  Serotype-15C -Erythromycin-S |  | 0 | 1
  Serotype-18C -Erythromycin-S |  | 0 | 1
  Serotype-19A -Erythromycin-S |  | 0 | 1
  Serotype-19F -Erythromycin-R |  | 0 | 1
  Serotype-19F -Erythromycin-S |  | 0 | 1
  Serotype-23F -Erythromycin-S |  | 0 | 1
  Serotype-N -Erythromycin-N |  | 1 | 4
  Serotype-4 -Tetracyclin-S |  | 0 | 1
  Serotype-6A -Tetracyclin-S |  | 0 | 1
  Serotype-6B -Tetracyclin-R |  | 0 | 4
  Serotype-6B -Tetracyclin-S |  | 0 | 2
  Serotype-7F -Tetracyclin-S |  | 1 | 1
  Serotype-14 -Tetracyclin-S |  | 0 | 5
  Serotype-15C -Tetracyclin-S |  | 0 | 1
  Serotype-18C -Tetracyclin-S |  | 0 | 1
  Serotype-19A -Tetracyclin-S |  | 0 | 1
  Serotype-19F -Tetracyclin-R |  | 0 | 1
  Serotype-19F -Tetracyclin-S |  | 0 | 1
  Serotype-23F -Tetracyclin-S |  | 0 | 1
  Serotype-N -Tetracyclin-N |  | 1 | 4
  Serotype-4 -Levoffloxacin-S |  | 0 | 1
  Serotype-6A -Levoffloxacin-S |  | 0 | 1
  Serotype-6B -Levoffloxacin-S |  | 0 | 6
  Serotype-7F -Levoffloxacin-S |  | 1 | 1
  Serotype-14 -Levoffloxacin-S |  | 0 | 5
  Serotype-15C -Levoffloxacin-S |  | 0 | 1
  Serotype-18C -Levoffloxacin-S |  | 0 | 1
  Serotype-19A -Levoffloxacin-S |  | 0 | 1
  Serotype-19F -Levoffloxacin-S |  | 0 | 2
  Serotype-23F -Levoffloxacin-S |  | 0 | 1
  Serotype-N -Levoffloxacin-N |  | 1 | 4
  Serotype-4 -Ceftriaxone-S |  | 0 | 1
  Serotype-6A -Ceftriaxone-S |  | 0 | 1
  Serotype-6B -Ceftriaxone-S |  | 0 | 6
  Serotype-7F -Ceftriaxone-S |  | 1 | 1
  Serotype-14 -Ceftriaxone-I |  | 0 | 1
  Serotype-14 -Ceftriaxone-S |  | 0 | 4
  Serotype-15C -Ceftriaxone-S |  | 0 | 1
  Serotype-18C -Ceftriaxone-S |  | 0 | 1
  Serotype-19A -Ceftriaxone-S |  | 0 | 1
  Serotype-19F -Ceftriaxone-S |  | 0 | 2
  Serotype-23F -Ceftriaxone-S |  | 0 | 1
  Serotype-N -Ceftriaxone-N |  | 1 | 4
  Serotype-4 -Clindamycin-S |  | 0 | 1
  Serotype-6A -Clindamycin-S |  | 0 | 1
  Serotype-6B -Clindamycin-R |  | 0 | 4
  Serotype-6B -Clindamycin-S |  | 0 | 2
  Serotype-7F -Clindamycin-S |  | 1 | 1
  Serotype-14 -Clindamycin-N |  | 0 | 1
  Serotype-14 -Clindamycin-S |  | 0 | 4
  Serotype-15C -Clindamycin-S |  | 0 | 1
  Serotype-18C -Clindamycin-S |  | 0 | 1
  Serotype-19A -Clindamycin-S |  | 0 | 1
  Serotype-19F -Clindamycin-R |  | 0 | 1
  Serotype-19F -Clindamycin-S |  | 0 | 1
  Serotype-23F -Clindamycin-S |  | 0 | 1
  Serotype-N -Clindamycin-N |  | 1 | 4

28. Secondary Outcome: Number of Subjects With Lower Respiratory Tract Infections (LRTIs) (in a Subset of Subjects in Turku Area )
Description: Analysis of this outcome was performed in the Turku area. The number of subjects reporting at least one LRTI any time after the administration of the first vaccine dose was tabulated.
Time Frame: From the administration of the first vaccine dose till the end of the blinded invasive disease (ID) Follow-up period (at least 30 months).
Population: The analysis was performed in a subset of vaccinated subjects including all vaccinated subjects enrolled in the 10PNPD-DIT-053 study in the Turku area and those vaccinated subjects enrolled in the 10PN-PD-DIT-043 study in the Turku area who agreed to take part in this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- 10Pn7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PNPD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 3689 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 7 to 11 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (7-11M Schedule). Refer to group description for 10Pn7-11M/053 Group for details on vaccine specifics and administration route in this group.
- Ctrl7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PNPD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 1812 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 7 to 11 months at enrolment. Subjects received the Engerix B (called also HBV) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (7-11M Schedule). Refer to group description for Ctrl7-11M/053 Group for details on vaccine specifics and administration route in this group.
- 10Pn12-18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PNPD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 6249 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 12 to 18 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for 10Pn12-18M/053 Group for details on vaccine specifics and administration route in this group.
- Ctrl12-18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PNPD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 3020 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 12 to 18 months at enrolment. Subjects received the Havrix (called also HAV) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for Ctrl12-18M/053 Group for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 243 | 190 | 171 | 31 | 22 | 62 | 48
Participants | 19 | 19 | 19 | 3 | 1 | 5 | 2

29. Secondary Outcome: Number of Subjects With Upper Respiratory Tract Infections (URTIs) (in a Subset of Subjects in Turku Area )
Description: Analysis of this outcome was performed in the Turku area. The number of subjects reporting at least one URTI any time after the administration of the first vaccine dose was tabulated.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 243 | 190 | 171 | 31 | 22 | 62 | 48
Participants | 158 | 124 | 94 | 14 | 15 | 27 | 19

30. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: Within 4 days (4D) after each vaccination (M0+4D, M1+4D [only for 3+1 schedule], M2+4D, M8+4D [booster dose] for 6W-6M subjects; M0+4D, M2+4D, M6+4D [booster dose] for 7M-11M subjects; M0+4D, M6+4D for 12M-18M subjects)
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 1846 | 1302 | 1066 | 852 | 237 | 202 | 363 | 270
Participants
  Any Pain, Dose 1 | 807 | 611 | 146 | 106 | 120 | 33 | 220 | 65
  Grade 3 Pain, Dose 1 | 60 | 43 | 2 | 3 | 6 | 0 | 19 | 0
  Any Redness (mm), Dose 1 | 936 | 675 | 270 | 214 | 137 | 48 | 203 | 93
  Grade 3 Redness (mm), Dose 1 | 56 | 48 | 3 | 0 | 17 | 0 | 39 | 0
  Any Swelling (mm), Dose 1 | 636 | 471 | 88 | 64 | 107 | 19 | 142 | 25
  Grade 3 Swelling (mm), Dose 1 | 89 | 69 | 4 | 1 | 20 | 9 | 35 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 1827 | 1287 | 1056 | 847 | 229 | 199 | 345 | 260
  Any Pain, Dose 2 | 662 | 509 | 114 | 94 | 108 | 38 | 242 | 78
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 1827 | 1287 | 1056 | 847 | 229 | 199 | 345 | 260
  Grade 3 Pain, Dose 2 | 23 | 28 | 2 | 1 | 11 | 0 | 45 | 0
  Any Redness (mm), Dose 2: number analyzed (Participants) | 1827 | 1287 | 1056 | 847 | 229 | 199 | 345 | 260
  Any Redness (mm), Dose 2 | 996 | 690 | 254 | 203 | 124 | 57 | 193 | 85
  Grade 3 Redness (mm), Dose 2: number analyzed (Participants) | 1827 | 1287 | 1056 | 847 | 229 | 199 | 345 | 260
  Grade 3 Redness (mm), Dose 2 | 48 | 63 | 3 | 0 | 21 | 0 | 49 | 1
  Any Swelling (mm), Dose 2: number analyzed (Participants) | 1827 | 1287 | 1056 | 847 | 229 | 199 | 345 | 260
  Any Swelling (mm), Dose 2 | 686 | 536 | 114 | 79 | 98 | 18 | 148 | 26
  Grade 3 Swelling (mm), Dose 2: number analyzed (Participants) | 1827 | 1287 | 1056 | 847 | 229 | 199 | 345 | 260
  Grade 3 Swelling (mm), Dose 2 | 67 | 91 | 4 | 1 | 19 | 0 | 34 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 3 | 538 |  | 102 |  |  |  |  |
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Grade 3 Pain, Dose 3 | 12 |  | 2 |  |  |  |  |
  Any Redness (mm), Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Any Redness (mm), Dose 3 | 963 |  | 300 |  |  |  |  |
  Grade 3 Redness (mm), Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Grade 3 Redness (mm), Dose 3 | 52 |  | 0 |  |  |  |  |
  Any Swelling (mm), Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Any Swelling (mm), Dose 3 | 676 |  | 144 |  |  |  |  |
  Grade 3 Swelling (mm), Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Grade 3 Swelling (mm), Dose 3 | 62 |  | 1 |  |  |  |  |
  Any Pain, Booster dose: number analyzed (Participants) | 1758 | 1258 | 1024 | 827 | 216 | 188 | 0 | 0
  Any Pain, Booster dose | 888 | 710 | 250 | 171 | 123 | 40 |  |
  Grade 3 Pain, Booster dose: number analyzed (Participants) | 1758 | 1258 | 1024 | 827 | 216 | 188 | 0 | 0
  Grade 3 Pain, Booster dose | 66 | 41 | 2 | 2 | 14 | 2 |  |
  Any Redness (mm), Booster dose: number analyzed (Participants) | 1758 | 1258 | 1024 | 827 | 216 | 188 | 0 | 0
  Any Redness (mm), Booster dose | 913 | 702 | 345 | 238 | 106 | 54 |  |
  Grade 3 Redness (mm), Booster dose: number analyzed (Participants) | 1758 | 1258 | 1024 | 827 | 216 | 188 | 0 | 0
  Grade 3 Redness (mm), Booster dose | 102 | 103 | 13 | 2 | 18 | 0 |  |
  Any Swelling (mm), Booster dose: number analyzed (Participants) | 1758 | 1258 | 1024 | 827 | 216 | 188 | 0 | 0
  Any Swelling (mm), Booster dose | 716 | 586 | 229 | 118 | 85 | 31 |  |
  Grade 3 Swelling (mm), Booster dose: number analyzed (Participants) | 1758 | 1258 | 1024 | 827 | 216 | 188 | 0 | 0
  Grade 3 Swelling (mm), Booster dose | 102 | 111 | 10 | 3 | 14 | 0 |  |

31. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were drowsiness, fever [defined as rectal temperature ≥ 38 degrees Celsius (°C) or oral/axillary/tympanic temperature equal to or above 37.5°C], irritability/fussiness and loss pf appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 fever = rectal temperature > 40°C. Grade 3 irritability/fussiness = cried that could not be comforted/prevented normal activity. Grade 3 loss of appetite = not eating at all. Related = a symptom assessed by investigator as causally related to the vaccination.
Time Frame: as for outcome 30
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 1846 | 1302 | 1066 | 852 | 237 | 202 | 363 | 270
Participants
  Any Drowsiness, Dose 1 | 1070 | 742 | 462 | 384 | 106 | 62 | 155 | 87
  Grade 3 Drowsiness, Dose 1 | 11 | 8 | 5 | 1 | 1 | 0 | 1 | 2
  Related Drowsiness, Dose 1 | 1054 | 738 | 453 | 374 | 103 | 57 | 152 | 81
  Any Temperature (Rectally)/(°C), Dose 1 | 388 | 289 | 82 | 78 | 38 | 16 | 74 | 28
  Grade 3 Temperature (Rectally)/(°C), Dose 1 | 2 | 0 | 1 | 0 | 8 | 0 | 2 | 2
  Related Temperature (Rectally)/(°C), Dose 1 | 381 | 284 | 78 | 74 | 35 | 13 | 69 | 25
  Any Irritability, Dose 1 | 1325 | 942 | 577 | 468 | 157 | 90 | 210 | 103
  Grade 3 Irritability, Dose 1 | 76 | 56 | 20 | 14 | 3 | 2 | 6 | 4
  Related Irritability, Dose 1 | 1298 | 937 | 565 | 460 | 157 | 83 | 201 | 96
  Any Loss of appetite, Dose 1 | 499 | 335 | 202 | 147 | 84 | 56 | 128 | 82
  Grade 3 Loss of appetite, Dose 1 | 1 | 3 | 2 | 0 | 0 | 1 | 2 | 4
  Related Loss of appetite, Dose 1 | 480 | 332 | 196 | 140 | 81 | 48 | 123 | 73
  Any Drowsiness, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Any Drowsiness, Dose 2 | 868 | 572 | 332 | 258 | 88 | 52 | 126 | 58
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Grade 3 Drowsiness, Dose 2 | 7 | 6 | 1 | 3 | 2 | 1 | 2 | 1
  Related Drowsiness, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Related Drowsiness, Dose 2 | 855 | 564 | 329 | 247 | 85 | 51 | 123 | 55
  Any Temperature (Rectally)/(°C), Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Any Temperature (Rectally)/(°C), Dose 2 | 380 | 382 | 78 | 80 | 44 | 20 | 55 | 11
  Grade 3 Temperature (Rectally)/(°C), Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Grade 3 Temperature (Rectally)/(°C), Dose 2 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1
  Related Temperature (Rectally)/(°C), Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Related Temperature (Rectally)/(°C), Dose 2 | 373 | 378 | 78 | 71 | 43 | 15 | 53 | 8
  Any Irritability, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Any Irritability, Dose 2 | 1254 | 822 | 532 | 408 | 139 | 94 | 193 | 72
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Grade 3 Irritability, Dose 2 | 73 | 44 | 13 | 14 | 7 | 1 | 3 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Related Irritability, Dose 2 | 1236 | 816 | 523 | 396 | 137 | 93 | 191 | 71
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Any Loss of appetite, Dose 2 | 434 | 323 | 187 | 149 | 69 | 56 | 109 | 57
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Grade 3 Loss of appetite, Dose 2 | 4 | 2 | 1 | 3 | 44 | 0 | 2 | 1
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 1828 | 1287 | 1056 | 847 | 229 | 198 | 345 | 260
  Related Loss of appetite, Dose 2 | 419 | 318 | 181 | 135 | 0 | 52 | 105 | 54
  Any Drowsiness, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Any Drowsiness, Dose 3 | 645 |  | 293 |  |  |  |  |
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 3 | 2 |  | 2 |  |  |  |  |
  Related Drowsiness, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 3 | 638 |  | 285 |  |  |  |  |
  Any Temperature (Rectally)/(°C), Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Any Temperature (Rectally)/(°C), Dose 3 | 347 |  | 110 |  |  |  |  |
  Grade 3 Temperature (Rectally)/(°C), Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Grade 3 Temperature (Rectally)/(°C), Dose 3 | 1 |  | 1 |  |  |  |  |
  Related Temperature (Rectally)/(°C), Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Related Temperature (Rectally)/(°C), Dose 3 | 336 |  | 106 |  |  |  |  |
  Any Irritability, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Any Irritability, Dose 3 | 1115 |  | 496 |  |  |  |  |
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Grade 3 Irritability, Dose 3 | 41 |  | 14 |  |  |  |  |
  Related Irritability, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Related Irritability, Dose 3 | 1100 |  | 492 |  |  |  |  |
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Any Loss of appetite, Dose 3 | 349 |  | 178 |  |  |  |  |
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Grade 3 Loss of appetite, Dose 3 | 3 |  | 0 |  |  |  |  |
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 1808 | 0 | 1052 | 0 | 0 | 0 | 0 | 0
  Related Loss of appetite, Dose 3 | 336 |  | 172 |  |  |  |  |
  Any Drowsiness, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Any Drowsiness, Booster dose | 721 | 561 | 307 | 243 | 92 | 47 |  |
  Grade 3 Drowsiness, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Grade 3 Drowsiness, Booster dose | 8 | 8 | 3 | 4 | 2 | 1 |  |
  Related Drowsiness, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Related Drowsiness, Booster dose | 699 | 548 | 300 | 233 | 87 | 46 |  |
  Any Temperature (Rectally)/(°C), Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Any Temperature (Rectally)/(°C), Booster dose | 391 | 333 | 142 | 120 | 42 | 11 |  |
  Grade 3 Temperature (Rectally)/(°C), Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Grade 3 Temperature (Rectally)/(°C), Booster dose | 3 | 0 | 0 | 1 | 1 | 0 |  |
  Related Temperature (Rectally)/(°C), Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Related Temperature (Rectally)/(°C), Booster dose | 371 | 319 | 134 | 110 | 41 | 8 |  |
  Any Irritability, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Any Irritability, Booster dose | 1124 | 816 | 491 | 410 | 129 | 84 |  |
  Grade 3 Irritability, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Grade 3 Irritability, Booster dose | 47 | 33 | 14 | 7 | 2 | 1 |  |
  Related Irritability, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Related Irritability, Booster dose | 1085 | 801 | 481 | 395 | 124 | 80 |  |
  Any Loss of appetite, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Any Loss of appetite, Booster dose | 549 | 411 | 260 | 186 | 64 | 46 |  |
  Grade 3 Loss of appetite, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Grade 3 Loss of appetite, Booster dose | 12 | 5 | 6 | 3 | 2 | 1 |  |
  Related Loss of appetite, Booster dose: number analyzed (Participants) | 1757 | 1257 | 1024 | 827 | 216 | 188 | 0 | 0
  Related Loss of appetite, Booster dose | 513 | 398 | 253 | 173 | 60 | 43 |  |

32. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (31D) after each vaccination (M0+31D, M1+31D [only for 3+1 schedule], M2+31D, M8+31D [booster dose] for 6W-6M subjects; M0+31D, M2+31D, M6+31D [booster dose] for 7M-11M subjects; M0+31D, M6+31D for 12M-18M subjects)
Population: Analysis was performed on the Total vaccinated cohort which included all subjects who had received at least one vaccination dose.
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 1849 | 1316 | 1069 | 859 | 241 | 204 | 368 | 271
Participants
  Unsolicited AEs, Primary vaccination | 1105 | 598 | 554 | 337 | 157 | 132 | 221 | 174
  Unsolicited AEs, Booster vaccination: number analyzed (Participants) | 1786 | 1275 | 1043 | 837 | 226 | 197 | 0 | 0
  Unsolicited AEs, Booster vaccination | 521 | 363 | 277 | 244 | 51 | 48 |  |

33. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: An event is defined as 'serious' when it meets one of the pre-defined outcomes described below: results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation; results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study subject. Medical or scientific judgement should be exercised in deciding whether reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalisation but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These should also be considered serious.
Time Frame: Following administration of the first vaccine dose up to study end (M0 up to M18 for subjects aged 6W to 6M at enrollment; M0 up to M16 for subjects aged 7M to 11M at enrollment; M0 up to M9 for subjects aged 12M to 18M at enrollment)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 1849 | 1316 | 1069 | 859 | 241 | 204 | 368 | 271
Participants | 163 | 96 | 77 | 74 | 24 | 18 | 23 | 14

34. Secondary Outcome: Number of Subjects Enrolled and Vaccinated in the 10PN-PD-DIT-043 and 10PN-PD-DIT-053 Study With Post-study SAEs Reported Via Passive Surveillance- Subjects Enrolled Aged 6 Weeks to 6 Months and 7 to 18 Months
Description: as for outcome 33
Time Frame: From the end of the blinded ID Follow-Up period (at least 30 months from the study start) up to the end of 18-month period after study unblinding
Population: Analysis was performed on the Total vaccinated cohort which included all subjects who had received at least one vaccination dose in the 10PN-PD-DIT-043 and 10PN-PD-DIT-053 study with post-study SAEs reported via passive surveillance.
Measure: Count of Participants; unit: Participants
Groups:
- 10Pn3+1-6W- 6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 8427 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (or 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule). Refer to group description for 10Pn3+1-6W-6M/053 Group for details on vaccine specifics and administration route in this group.
- 10Pn2+1-6W- 6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 9112 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (or 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group description for 10Pn2+1-6W-6M/053 Group for details on vaccine specifics and administration route in this group.
- Ctrl-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 8872 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B-thio free vaccine (or HBV vaccine) according to either a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule), or according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group descriptions for Ctrl3+1-6W-6M/053 and Ctrl2+1-6W-6M/053 groups for details on vaccine specifics and administration route in this group.
- 10Pn7- 11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 3689 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 7 to 11 months at enrolment. Subjects received the Synflorix (or 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (7-11M Schedule). Refer to group description for 10Pn7-11M/053 Group for details on vaccine specifics and administration route in this group.
- Ctrl7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 1812 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 7 to 11 months at enrolment. Subjects received the Engerix B-thio free (or HBV) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months 1908 since the previous vaccine dose (minimum 4 months) (7-11M Schedule). Refer to group description for Ctrl7-11M/053 Group for details on vaccine specifics and administration route in this group.
- 10Pn12- 18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 6249 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 12 to 18 months at enrolment. Subjects received the Synflorix (or 10Pn-PD-DiT, or 10Pn or GSK1024850A) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for 10Pn12-18M/053 Group for details on vaccine specifics and administration route in this group.
- Ctrl12-18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) (i.e. 3020 subjects) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 12 to 18 months at enrolment. Subjects received the Synflorix (or 10Pn-PD-DiT, or 10Pn) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for Ctrl12-18M/053 Group for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn3+1-6W- 6M/043+053 Group | 10Pn2+1-6W- 6M/043+053 Group | Ctrl-6W-6M/043+053 Group | 10Pn7- 11M/043+053 Group | Ctrl7-11M/043+053 Group | 10Pn12- 18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 10273 | 10054 | 10201 | 3880 | 1908 | 6535 | 3126
Participants | 1 | 2 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STREPTOCOCCUS PNEUMONIAE PATHOGENS (S. PN.), ANY PATHOGEN. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of swabs associated with the specified bacteria was tabulated. The "prior to dose 1" nasopharyngeal swab samples collected from subjects within their first 7 months of age were obtained solely from the Immuno subset (The Immuno subset was constituted of the first +/- 1500 subjects from whom blood samples were collected, according to age and treatment groups).
Time Frame: At 3 months (mths) of age (prior to dose 1); at 6 mths of age (1 mth post dose 3 or post dose 2); at 11-12 mths of age (pre-booster dose); at 14-15 mths of age (3 mths post-booster); at 18-22 mths of age (10 mths post-booster)
Population: The Total Vaccinated cohort for analysis of carriage included all vaccinated subjects for whom data concerning carriage outcome measures were available.
Measure: Number; unit: swab samples
Groups:
- Ctrl-6W-6M/053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) studies and aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B-thio free vaccine (or HBV vaccine) according to either a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule), or according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group descriptions for Ctrl3+1-6W-6M/053 and Ctrl2+1-6W-6M/053 groups for details on vaccine specifics and administration route in this group.
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1803 | 1289 | 1897
swab samples
  3 Months: number analyzed (Participants) | 253 | 253 | 341
  3 Months | 49 | 31 | 56
  6 Months | 412 | 323 | 464
  11-12 Months: number analyzed (Participants) | 1784 | 1269 | 1877
  11-12 Months | 500 | 383 | 604
  14-15 Months: number analyzed (Participants) | 1727 | 1227 | 1814
  14-15 Months | 512 | 370 | 638
  18-22 Months: number analyzed (Participants) | 1686 | 1216 | 1769
  18-22 Months | 503 | 430 | 736

36. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STREPTOCOCCUS PNEUMONIAE PATHOGENS (S. PN.), ANY PATHOGEN. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of swabs associated with the specified bacteria was tabulated.
Time Frame: At 7-11 months (mths) of age (prior to dose 1); at 9-13 mths of age (1 mth post dose 2); at 13-17 mths of age (pre-booster dose); at 16-20 mths of age (3 mths post-booster); at 23-27 mths of age (10 mths post-booster)
Population: as for outcome 35
Measure: Number; unit: swab samples
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 236 | 200
swab samples
  7-11 Months: number analyzed (Participants) | 236 | 198
  7-11 Months | 69 | 58
  9-13 Months: number analyzed (Participants) | 230 | 200
  9-13 Months | 79 | 56
  13-17 Months: number analyzed (Participants) | 225 | 197
  13-17 Months | 81 | 87
  16-20 Months: number analyzed (Participants) | 209 | 179
  16-20 Months | 75 | 72
  23-27 Months: number analyzed (Participants) | 200 | 175
  23-27 Months | 68 | 75

37. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STREPTOCOCCUS PNEUMONIAE PATHOGENS (S. PN.), ANY PATHOGEN. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: At 12-18 months (mths) of age (prior to dose 1); at 19-25 mths of age (1 mth post dose 2); at 21-27 mths of age (3 months post dose 2)
Population: as for outcome 35
Measure: Number; unit: swab samples
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 358 | 265
swab samples
  12-18 Months | 125 | 88
  19-25 Months: number analyzed (Participants) | 340 | 255
  19-25 Months | 152 | 112
  21-27 Months: number analyzed (Participants) | 338 | 254
  21-27 Months | 132 | 105

38. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STREPTOCOCCUS PNEUMONIAE (S. PN.) VACCINE SEROTYPES. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of swabs associated with the specified bacteria was tabulated. The "prior to dose 1" nasopharyngeal swab samples collected from subjects within their first 7 months of age were obtained solely from the Immuno subset (The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups).
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Number; unit: swab samples
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1803 | 1289 | 1897
swab samples
  3 Months: number analyzed (Participants) | 253 | 253 | 341
  3 Months | 29 | 18 | 30
  6 Months | 183 | 159 | 237
  11-12 Months: number analyzed (Participants) | 1784 | 1269 | 1877
  11-12 Months | 229 | 178 | 342
  14-15 Months: number analyzed (Participants) | 1727 | 1227 | 1814
  14-15 Months | 209 | 153 | 364
  18-22 Months: number analyzed (Participants) | 1686 | 1216 | 1769
  18-22 Months | 169 | 176 | 404

39. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STREPTOCOCCUS PNEUMONIAE (S. PN.) VACCINE SEROTYPES. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 35
Measure: Number; unit: swab samples
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 236 | 200
swab samples
  7-11 Months: number analyzed (Participants) | 236 | 198
  7-11 Months | 44 | 34
  9-13 Months: number analyzed (Participants) | 230 | 200
  9-13 Months | 43 | 35
  13-17 Months: number analyzed (Participants) | 225 | 197
  13-17 Months | 43 | 55
  16-20 Months: number analyzed (Participants) | 209 | 179
  16-20 Months | 34 | 47
  23-27 Months: number analyzed (Participants) | 200 | 175
  23-27 Months | 28 | 48

40. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STREPTOCOCCUS PNEUMONIAE (S. PN.) VACCINE SEROTYPES. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: as for outcome 37
Population: as for outcome 35
Measure: Number; unit: swab samples
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 358 | 265
swab samples
  12-18 Months | 70 | 57
  19-25 Months: number analyzed (Participants) | 340 | 255
  19-25 Months | 69 | 70
  21-27 Months: number analyzed (Participants) | 338 | 254
  21-27 Months | 64 | 53

41. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW STREPTOCOCCUS PNEUMONIAE (S. PN.) STRAINS, ANY PATHOGEN, IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of subjects with new acquisition associated to the specified bacteria at the considered time point was tabulated.
Time Frame: At 11-12 mths of age (pre-booster dose); at 14-15 mths of age (3 mths post-booster); at 18-22 mths of age (10 mths post-booster)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1780 | 1269 | 1874
Participants
  11-12 Months | 331 | 246 | 415
  14-15 Months: number analyzed (Participants) | 1723 | 1222 | 1807
  14-15 Months | 562 | 400 | 692
  18-22 Months: number analyzed (Participants) | 1675 | 1200 | 1752
  18-22 Months | 818 | 609 | 1023

42. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW STREPTOCOCCUS PNEUMONIAE (S. PN.) STRAINS, ANY PATHOGEN, IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 41
Time Frame: At 9-13 mths of age (1 mth post dose 2); at 13-17 mths of age (pre-booster dose); at 16-20 mths of age (3 mths post-booster); at 23-27 mths of age (10 mths post-booster)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 226 | 195
Participants
  9-13 Months | 36 | 30
  13-17 Months: number analyzed (Participants) | 221 | 192
  13-17 Months | 78 | 83
  16-20 Months: number analyzed (Participants) | 205 | 175
  16-20 Months | 95 | 100
  23-27 Months: number analyzed (Participants) | 194 | 170
  23-27 Months | 117 | 116

43. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW STREPTOCOCCUS PNEUMONIAE (S. PN.) STRAINS, ANY PATHOGEN, IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 41
Time Frame: At 19-25 mths of age (1 mth post dose 2); at 21-27 mths of age (3 months post dose 2)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 333 | 249
Participants
  19-25 Months | 130 | 94
  21-27 Months: number analyzed (Participants) | 330 | 246
  21-27 Months | 166 | 133

44. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW STREPTOCOCCUS PNEUMONIAE (S. PN.) VACCINE SEROTYPE STRAINS, IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: as for outcome 41
Time Frame: as for outcome 41
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1780 | 1269 | 1874
Participants
  11-12 Months | 131 | 97 | 223
  14-15 Months: number analyzed (Participants) | 1723 | 1222 | 1807
  14-15 Months | 221 | 156 | 387
  18-22 Months: number analyzed (Participants) | 1675 | 1200 | 1752
  18-22 Months | 326 | 269 | 626

45. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW STREPTOCOCCUS PNEUMONIAE (S. PN.) VACCINE SEROTYPE STRAINS, IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 41
Time Frame: as for outcome 42
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 226 | 195
Participants
  9-13 Months | 18 | 17
  13-17 Months: number analyzed (Participants) | 221 | 192
  13-17 Months | 41 | 51
  16-20 Months: number analyzed (Participants) | 205 | 175
  16-20 Months | 50 | 70
  23-27 Months: number analyzed (Participants) | 194 | 170
  23-27 Months | 62 | 88

46. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW STREPTOCOCCUS PNEUMONIAE (S. PN.) VACCINE SEROTYPE STRAINS, IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 41
Time Frame: At 19-25 mths of age (1 mth post dose 2); at 21-27 mths of age (3 months post dose 2)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 333 | 249
Participants
  19-25 Months | 53 | 55
  21-27 Months: number analyzed (Participants) | 330 | 246
  21-27 Months | 78 | 74

47. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH HAEMOPHILUS INFLUENZAE (H. INFL.) PATHOGENS. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of swabs associated with the specified bacteria was tabulated. The "prior to dose 1" nasopharyngeal swab samples collected from subjects within their first 7 months of age were obtained solely from the Immuno subset (The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups). Data presented only include results from samples confirmed as positive for Hi/NTHi after differentiation from H. haemolyticus by PCR assay.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1803 | 1289 | 1897
Swab samples
  3 Months: number analyzed (Participants) | 253 | 253 | 341
  3 Months | 6 | 4 | 10
  6 Months | 57 | 36 | 46
  11-12 Months: number analyzed (Participants) | 1784 | 1269 | 1877
  11-12 Months | 84 | 72 | 87
  14-15 Months: number analyzed (Participants) | 1726 | 1227 | 1814
  14-15 Months | 121 | 84 | 92
  18-22 Months: number analyzed (Participants) | 1684 | 1212 | 1768
  18-22 Months | 211 | 128 | 190

48. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH HAEMOPHILUS INFLUENZAE (H. INFL.) PATHOGENS. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of swabs associated with the specified bacteria was tabulated. Data presented only include results from samples confirmed as positive for Hi /NTHi after differentiation from H. haemolyticus by PCR assay.
Time Frame: as for outcome 36
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 236 | 200
Swab samples
  7-11 Months: number analyzed (Participants) | 236 | 198
  7-11 Months | 6 | 8
  9-13 Months: number analyzed (Participants) | 230 | 200
  9-13 Months | 8 | 9
  13-17 Months: number analyzed (Participants) | 225 | 197
  13-17 Months | 22 | 14
  16-20 Months: number analyzed (Participants) | 209 | 179
  16-20 Months | 17 | 13
  23-27 Months: number analyzed (Participants) | 200 | 175
  23-27 Months | 21 | 15

49. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH HAEMOPHILUS INFLUENZAE (H. INFL.) PATHOGENS. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of swabs associated with the specified bacteria was tabulated. Data presented only include results from samples confirmed as positive for Hi/NTHi after differentiation from H. haemolyticus by PCR assay.
Time Frame: as for outcome 37
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 358 | 265
Swab samples
  12-18 Months | 21 | 12
  19-25 Months: number analyzed (Participants) | 340 | 255
  19-25 Months | 24 | 21
  21-27 Months: number analyzed (Participants) | 338 | 254
  21-27 Months | 27 | 29

50. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW HAEMOPHILUS INFLUENZAE (H. INFL.) PATHOGENS IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of subjects with new acquisition associated to the specified bacteria at the considered time point was tabulated. Data presented only include results from samples confirmed as positive for Hi/NTHi after differentiation from H. haemolyticus by PCR assay.
Time Frame: At 11-12 mths of age (pre-booster dose) ; at 14-15 mths of age ( 3 mths post-booster) ; at 18-22 mths of age (10 mths post-booster)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1780 | 1269 | 1874
Participants
  11-12 Months | 77 | 65 | 83
  14-15 Months: number analyzed (Participants) | 1722 | 1222 | 1807
  14-15 Months | 176 | 139 | 157
  18-22 Months: number analyzed (Participants) | 1672 | 1196 | 1751
  18-22 Months | 349 | 240 | 313

51. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW HAEMOPHILUS INFLUENZAE (H. INFL.) PATHOGENS IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 50
Time Frame: At 9-13 mths of age (1 mth post dose 2); at 13-17 mths of age (pre-booster dose); at 16-20 mths of age (3 mths post-booster) at 23-27 mths of age (10 mths post-booster)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 226 | 195
Participants
  9-13 Months | 8 | 9
  13-17 Months: number analyzed (Participants) | 221 | 192
  13-17 Months | 29 | 19
  16-20 Months: number analyzed (Participants) | 205 | 175
  16-20 Months | 37 | 28
  23-27 Months: number analyzed (Participants) | 194 | 170
  23-27 Months | 55 | 39

52. Secondary Outcome: NUMBER OF SUBJECTS WITH ACQUISITION OF NEW HAEMOPHILUS INFLUENZAE (H. INFL.) PATHOGENS IDENTIFIED IN NASOPHARYNGEAL SWABS. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 50
Time Frame: At 19-25 mths of age (1 mth post dose 2); at 21-27 mths of age (3 months post dose 2)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 333 | 249
Participants
  19-25 Months | 19 | 20
  21-27 Months: number analyzed (Participants) | 330 | 246
  21-27 Months | 37 | 41

53. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH MORAXELLA CATARRHALIS PATHOGENS. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: At each time point where a swab sample result was available, the number/percentage of swabs associated with the specified bacteria was tabulated. The "prior to dose 1" nasopharyngeal swab samples collected from subjects within their first 7 months of age were obtained solely from the Immuno subset (The Immuno subset was constituted of the first 1500 subjects from whom blood samples were collected, according to age and treatment groups).
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1803 | 1289 | 1897
Swab samples
  3 Months: number analyzed (Participants) | 253 | 253 | 341
  3 Months | 57 | 58 | 76
  6 Months | 459 | 345 | 486
  11-12 Months: number analyzed (Participants) | 1784 | 1269 | 1877
  11-12 Months | 671 | 493 | 733
  14-15 Months: number analyzed (Participants) | 1727 | 1227 | 1814
  14-15 Months | 612 | 466 | 668
  18-22 Months: number analyzed (Participants) | 1686 | 1216 | 1769
  18-22 Months | 794 | 566 | 780

54. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH MORAXELLA CATARRHALIS PATHOGENS. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: At 7-11 months (mths) of age (prior to dose 1); at 9-13 mths of age (1 mth post dose 2) ; at 13-17 mths of age (pre-booster dose) ; at 16-20 mths of age ( 3 mths post-booster) ; at 23-27 mths of age (10 mths post-booster)
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 236 | 200
Swab samples
  7-11 Months: number analyzed (Participants) | 236 | 198
  7-11 Months | 69 | 59
  9-13 Months: number analyzed (Participants) | 230 | 200
  9-13 Months | 73 | 61
  13-17 Months: number analyzed (Participants) | 225 | 197
  13-17 Months | 109 | 98
  16-20 Months: number analyzed (Participants) | 209 | 179
  16-20 Months | 91 | 81
  23-27 Months: number analyzed (Participants) | 200 | 175
  23-27 Months | 83 | 63

55. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH MORAXELLA CATARRHALIS PATHOGENS. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: as for outcome 37
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 358 | 265
Swab samples
  12-18 Months | 143 | 72
  19-25 Months: number analyzed (Participants) | 340 | 255
  19-25 Months | 167 | 129
  21-27 Months: number analyzed (Participants) | 338 | 254
  21-27 Months | 143 | 120

56. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH GROUP A STREPTOCOCCUS PATHOGENS. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: as for outcome 38
Time Frame: At 3 months (mths) of age (prior to dose 1); at 6 mths of age (1 mth post dose 3 or post dose 2) ; at 11-12 mths of age (pre-booster dose) ; at 14-15 mths of age ( 3 mths post-booster) ; at 18-22 mths of age (10 mths post-booster)
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1803 | 1289 | 1897
Swab samples
  3 Months: number analyzed (Participants) | 253 | 253 | 341
  3 Months | 0 | 0 | 1
  6 Months | 10 | 5 | 8
  11-12 Months: number analyzed (Participants) | 1784 | 1269 | 1877
  11-12 Months | 9 | 8 | 5
  14-15 Months: number analyzed (Participants) | 1727 | 1227 | 1814
  14-15 Months | 4 | 5 | 10
  18-22 Months: number analyzed (Participants) | 1686 | 1216 | 1769
  18-22 Months | 5 | 5 | 7

57. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH GROUP A STREPTOCOCCUS PATHOGENS. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: as for outcome 54
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 236 | 200
Swab samples
  7-11 Months: number analyzed (Participants) | 236 | 198
  7-11 Months | 1 | 1
  9-13 Months: number analyzed (Participants) | 230 | 200
  9-13 Months | 0 | 3
  13-17 Months: number analyzed (Participants) | 225 | 197
  13-17 Months | 0 | 1
  16-20 Months: number analyzed (Participants) | 209 | 179
  16-20 Months | 0 | 2
  23-27 Months: number analyzed (Participants) | 200 | 175
  23-27 Months | 2 | 1

58. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH GROUP A STREPTOCOCCUS PATHOGENS. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: as for outcome 37
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 358 | 265
Swab samples
  12-18 Months | 3 | 0
  19-25 Months: number analyzed (Participants) | 340 | 255
  19-25 Months | 2 | 0
  21-27 Months: number analyzed (Participants) | 338 | 254
  21-27 Months | 0 | 2

59. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STAPHYLOCOCCUS AUREUS PATHOGENS. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: as for outcome 38
Time Frame: as for outcome 56
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1803 | 1289 | 1897
Swab samples
  3 Months: number analyzed (Participants) | 253 | 253 | 341
  3 Months | 111 | 108 | 144
  6 Months | 762 | 515 | 796
  11-12 Months: number analyzed (Participants) | 1784 | 1269 | 1877
  11-12 Months | 468 | 306 | 462
  14-15 Months: number analyzed (Participants) | 1727 | 1227 | 1814
  14-15 Months | 387 | 282 | 373
  18-22 Months: number analyzed (Participants) | 1686 | 1216 | 1769
  18-22 Months | 255 | 182 | 266

60. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STAPHYLOCOCCUS AUREUS PATHOGENS. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: as for outcome 54
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 236 | 200
Swab samples
  7-11 Months: number analyzed (Participants) | 236 | 198
  7-11 Months | 60 | 53
  9-13 Months: number analyzed (Participants) | 230 | 200
  9-13 Months | 53 | 63
  13-17 Months: number analyzed (Participants) | 225 | 197
  13-17 Months | 32 | 26
  16-20 Months: number analyzed (Participants) | 209 | 179
  16-20 Months | 34 | 31
  23-27 Months: number analyzed (Participants) | 200 | 175
  23-27 Months | 30 | 36

61. Secondary Outcome: NUMBER OF NASOPHARYNGEAL SWABS WITH STAPHYLOCOCCUS AUREUS PATHOGENS. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 36
Time Frame: as for outcome 37
Population: as for outcome 35
Measure: Number; unit: Swab samples
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 358 | 265
Swab samples
  12-18 Months | 45 | 38
  19-25 Months: number analyzed (Participants) | 340 | 255
  19-25 Months | 47 | 41
  21-27 Months: number analyzed (Participants) | 338 | 254
  21-27 Months | 39 | 40

62. Secondary Outcome: PNEUMOCOCCAL ANTIBODY CONCENTRATIONS AGAINST PNEUMOCOCCAL VACCINE SEROTYPES, IN THE IMMUNO SUBSET, IN SUBJECTS RECEIVING 3+1 INFANT SCHEDULES OF 10PN
Description: Antibody concentrations were measured by 22F -inhibition enzyme-linked Immunosorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). Serotypes assessed were the pneumococcal vaccine serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The cut-off of the assay was >= 0.05 µg/mL. The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups.
Time Frame: At 6 mths of age (1 mth post dose 3); at 11-12 mths of age (pre-booster dose) ; at 12-13 mths of age ( 1 mth post-booster) ; at 18-22 mths of age (10 mths post-booster)
Population: The According-to-Protocol cohort for immunogenicity included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn3+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group
Number analyzed (Participants) | 209 | 123
µg/mL
  ANTI-1, 6 months: number analyzed (Participants) | 208 | 121
  ANTI-1, 6 months | 1.86 [1.68 to 2.05] | 0.03 [0.03 to 0.04]
  ANTI-1, 11-12 months: number analyzed (Participants) | 202 | 122
  ANTI-1, 11-12 months | 0.54 [0.48 to 0.61] | 0.03 [0.03 to 0.03]
  ANTI-1, 12-13 months: number analyzed (Participants) | 189 | 119
  ANTI-1, 12-13 months | 2.13 [1.88 to 2.41] | 0.03 [0.03 to 0.04]
  ANTI-1, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-1, 18-22 months | 0.50 [0.44 to 0.57] | 0.04 [0.04 to 0.05]
  ANTI-4, 6 months: number analyzed (Participants) | 208 | 122
  ANTI-4, 6 months | 2.47 [2.23 to 2.75] | 0.03 [0.03 to 0.03]
  ANTI-4, 11-12 months: number analyzed (Participants) | 203 | 122
  ANTI-4, 11-12 months | 0.97 [0.86 to 1.09] | 0.03 [0.03 to 0.03]
  ANTI-4, 12-13: number analyzed (Participants) | 189 | 116
  ANTI-4, 12-13 | 3.61 [3.20 to 4.06] | 0.03 [0.03 to 0.03]
  ANTI-4, 18-22: number analyzed (Participants) | 185 | 113
  ANTI-4, 18-22 | 0.62 [0.54 to 0.71] | 0.03 [0.03 to 0.03]
  ANTI-5, 6 months: number analyzed (Participants) | 208 | 121
  ANTI-5, 6 months | 2.73 [2.47 to 3.01] | 0.03 [0.03 to 0.03]
  ANTI-5, 11-12 months: number analyzed (Participants) | 201 | 123
  ANTI-5, 11-12 months | 1.07 [0.95 to 1.19] | 0.04 [0.04 to 0.05]
  ANTI-5, 12-13: number analyzed (Participants) | 189 | 120
  ANTI-5, 12-13 | 3.27 [2.87 to 3.73] | 0.05 [0.04 to 0.06]
  ANTI-5, 18-22: number analyzed (Participants) | 185 | 113
  ANTI-5, 18-22 | 0.85 [0.75 to 0.97] | 0.10 [0.08 to 0.13]
  ANTI-6B, 6 months: number analyzed (Participants) | 208 | 122
  ANTI-6B, 6 months | 0.51 [0.43 to 0.62] | 0.03 [0.03 to 0.03]
  ANTI-6B, 11-12 months: number analyzed (Participants) | 203 | 123
  ANTI-6B, 11-12 months | 0.58 [0.50 to 0.67] | 0.03 [0.03 to 0.03]
  ANTI-6B, 12-13: number analyzed (Participants) | 189 | 120
  ANTI-6B, 12-13 | 1.43 [1.22 to 1.68] | 0.03 [0.03 to 0.03]
  ANTI-6B, 18-22: number analyzed (Participants) | 185 | 113
  ANTI-6B, 18-22 | 0.60 [0.50 to 0.72] | 0.04 [0.04 to 0.05]
  ANTI-7F, 6 months: number analyzed (Participants) | 209 | 120
  ANTI-7F, 6 months | 2.90 [2.62 to 3.20] | 0.03 [0.03 to 0.04]
  ANTI-7F, 11-12 months: number analyzed (Participants) | 202 | 122
  ANTI-7F, 11-12 months | 1.56 [1.40 to 1.74] | 0.04 [0.03 to 0.04]
  ANTI-7F, 12-13 months: number analyzed (Participants) | 189 | 120
  ANTI-7F, 12-13 months | 4.25 [3.80 to 4.75] | 0.04 [0.03 to 0.04]
  ANTI-7F, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-7F, 18-22 months | 1.19 [1.07 to 1.32] | 0.05 [0.04 to 0.05]
  ANTI-9V, 6 months: number analyzed (Participants) | 208 | 122
  ANTI-9V, 6 months | 2.23 [2.00 to 2.48] | 0.03 [0.03 to 0.03]
  ANTI-9V, 11-12 months: number analyzed (Participants) | 203 | 121
  ANTI-9V, 11-12 months | 1.35 [1.20 to 1.51] | 0.03 [0.03 to 0.03]
  ANTI-9V, 12-13 months: number analyzed (Participants) | 188 | 119
  ANTI-9V, 12-13 months | 3.98 [3.56 to 4.46] | 0.03 [0.03 to 0.03]
  ANTI-9V, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-9V, 18-22 months | 1.32 [1.16 to 1.50] | 0.03 [0.03 to 0.04]
  ANTI-14, 6 months: number analyzed (Participants) | 209 | 121
  ANTI-14, 6 months | 5.00 [4.46 to 5.61] | 0.07 [0.06 to 0.09]
  ANTI-14, 11-12 months: number analyzed (Participants) | 202 | 121
  ANTI-14, 11-12 months | 2.52 [2.19 to 2.91] | 0.05 [0.04 to 0.06]
  ANTI-14, 12-13 months: number analyzed (Participants) | 189 | 118
  ANTI-14, 12-13 months | 6.40 [5.62 to 7.29] | 0.06 [0.05 to 0.07]
  ANTI-14, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-14, 18-22 months | 1.98 [1.70 to 2.30] | 0.08 [0.06 to 0.11]
  ANTI-18C, 6 months: number analyzed (Participants) | 209 | 121
  ANTI-18C, 6 months | 6.51 [5.63 to 7.54] | 0.03 [0.03 to 0.04]
  ANTI-18C, 11-12 months: number analyzed (Participants) | 202 | 123
  ANTI-18C, 11-12 months | 2.45 [2.10 to 2.86] | 0.03 [0.03 to 0.03]
  ANTI-18C, 12-13 months: number analyzed (Participants) | 189 | 119
  ANTI-18C, 12-13 months | 10.43 [8.94 to 12.18] | 0.03 [0.03 to 0.03]
  ANTI-18C, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-18C, 18-22 months | 2.18 [1.89 to 2.53] | 0.04 [0.03 to 0.04]
  ANTI-19F, 6 months: number analyzed (Participants) | 209 | 122
  ANTI-19F, 6 months | 5.91 [5.06 to 6.89] | 0.06 [0.05 to 0.07]
  ANTI-19F, 11-12 months: number analyzed (Participants) | 202 | 122
  ANTI-19F, 11-12 months | 2.73 [2.36 to 3.16] | 0.05 [0.04 to 0.06]
  ANTI-19F, 12-13 months: number analyzed (Participants) | 189 | 116
  ANTI-19F, 12-13 months | 8.04 [7.04 to 9.17] | 0.04 [0.03 to 0.05]
  ANTI-19F, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-19F, 18-22 months | 2.17 [1.84 to 2.55] | 0.07 [0.05 to 0.08]
  ANTI-23F, 6 months: number analyzed (Participants) | 208 | 121
  ANTI-23F, 6 months | 0.68 [0.56 to 0.83] | 0.03 [0.03 to 0.03]
  ANTI-23F, 11-12 months: number analyzed (Participants) | 202 | 121
  ANTI-23F, 11-12 months | 0.73 [0.62 to 0.87] | 0.03 [0.03 to 0.03]
  ANTI-23F, 12-13 months: number analyzed (Participants) | 189 | 119
  ANTI-23F, 12-13 months | 2.30 [1.90 to 2.77] | 0.03 [0.03 to 0.04]
  ANTI-23F, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-23F, 18-22 months | 0.95 [0.79 to 1.13] | 0.05 [0.04 to 0.06]

63. Secondary Outcome: PNEUMOCOCCAL ANTIBODY CONCENTRATIONS AGAINST PNEUMOCOCCAL VACCINE SEROTYPES, IN THE IMMUNO SUBSET, IN SUBJECTS RECEIVING 2+1 INFANT SCHEDULES OF 10PN
Description: Antibody concentrations were measured by 22F-inhibition enzyme-linked Immunosorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). Serotypes assessed were the pneumococcal vaccine serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The cut-off of the assay was >= 0.05 µg/mL. The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups.
Time Frame: At 6 mths of age (1 mth post dose 2); at 11-12 mths of age (pre-booster dose) ; at 12-13 mths of age ( 1 mth post-booster) ; at 18-22 mths of age (10 mths post-booster)
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn2+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group
Number analyzed (Participants) | 209 | 142
µg/mL
  ANTI-1, 6 months: number analyzed (Participants) | 205 | 142
  ANTI-1, 6 months | 1.37 [1.25 to 1.52] | 0.03 [0.03 to 0.03]
  ANTI-1, 11-12 months: number analyzed (Participants) | 209 | 132
  ANTI-1, 11-12 months | 0.42 [0.37 to 0.47] | 0.03 [0.03 to 0.04]
  ANTI-1, 12-13 months: number analyzed (Participants) | 193 | 127
  ANTI-1, 12-13 months | 1.91 [1.72 to 2.12] | 0.04 [0.03 to 0.04]
  ANTI-1, 18-22 months: number analyzed (Participants) | 189 | 122
  ANTI-1, 18-22 months | 0.36 [0.32 to 0.40] | 0.05 [0.04 to 0.06]
  ANTI-4, 6 months: number analyzed (Participants) | 204 | 141
  ANTI-4, 6 months | 1.87 [1.68 to 2.07] | 0.03 [0.03 to 0.03]
  ANTI-4, 11-12 months: number analyzed (Participants) | 209 | 134
  ANTI-4, 11-12 months | 0.72 [0.64 to 0.81] | 0.03 [0.03 to 0.03]
  ANTI-4, 12-13 months: number analyzed (Participants) | 193 | 125
  ANTI-4, 12-13 months | 3.16 [2.84 to 3.52] | 0.03 [0.03 to 0.04]
  ANTI-4, 18-22 months: number analyzed (Participants) | 189 | 122
  ANTI-4, 18-22 months | 0.59 [0.52 to 0.67] | 0.03 [0.03 to 0.04]
  ANTI-5, 6 months: number analyzed (Participants) | 204 | 139
  ANTI-5, 6 months | 1.97 [1.76 to 2.19] | 0.03 [0.03 to 0.04]
  ANTI-5, 11-12 months: number analyzed (Participants) | 209 | 133
  ANTI-5, 11-12 months | 0.71 [0.63 to 0.80] | 0.04 [0.04 to 0.05]
  ANTI-5, 12-13 months: number analyzed (Participants) | 193 | 128
  ANTI-5, 12-13 months | 2.82 [2.52 to 3.15] | 0.06 [0.05 to 0.08]
  ANTI-5, 18-22 months: number analyzed (Participants) | 189 | 122
  ANTI-5, 18-22 months | 0.83 [0.73 to 0.94] | 0.09 [0.08 to 0.11]
  ANTI-6B, 6 months: number analyzed (Participants) | 205 | 142
  ANTI-6B, 6 months | 0.32 [0.27 to 0.37] | 0.03 [0.03 to 0.03]
  ANTI-6B, 11-12 months: number analyzed (Participants) | 209 | 133
  ANTI-6B, 11-12 months | 0.42 [0.36 to 0.48] | 0.03 [0.03 to 0.03]
  ANTI-6B, 12-13 months: number analyzed (Participants) | 193 | 127
  ANTI-6B, 12-13 months | 1.43 [1.25 to 1.65] | 0.03 [0.03 to 0.04]
  ANTI-6B, 18-22 months: number analyzed (Participants) | 189 | 124
  ANTI-6B, 18-22 months | 0.58 [0.48 to 0.70] | 0.06 [0.05 to 0.07]
  ANTI-7F, 6 months: number analyzed (Participants) | 205 | 140
  ANTI-7F, 6 months | 1.76 [1.57 to 1.97] | 0.03 [0.03 to 0.04]
  ANTI-7F, 11-12 months: number analyzed (Participants) | 209 | 132
  ANTI-7F, 11-12 months | 0.96 [0.86 to 1.07] | 0.03 [0.03 to 0.04]
  ANTI-7F, 12-13 months: number analyzed (Participants) | 193 | 129
  ANTI-7F, 12-13 months | 3.62 [3.28 to 4.01] | 0.03 [0.03 to 0.04]
  ANTI-7F, 18-22 months: number analyzed (Participants) | 189 | 122
  ANTI-7F, 18-22 months | 1.27 [1.15 to 1.41] | 0.04 [0.04 to 0.05]
  ANTI-9V, 6 months: number analyzed (Participants) | 205 | 140
  ANTI-9V, 6 months | 1.38 [1.24 to 1.54] | 0.03 [0.03 to 0.03]
  ANTI-9V, 11-12 months: number analyzed (Participants) | 209 | 133
  ANTI-9V, 11-12 months | 0.87 [0.77 to 0.97] | 0.03 [0.03 to 0.03]
  ANTI-9V, 12-13 months: number analyzed (Participants) | 193 | 127
  ANTI-9V, 12-13 months | 3.88 [3.47 to 4.33] | 0.03 [0.03 to 0.03]
  ANTI-9V, 18-22 months: number analyzed (Participants) | 189 | 122
  ANTI-9V, 18-22 months | 0.92 [0.82 to 1.03] | 0.04 [0.03 to 0.04]
  ANTI-14, 6 months: number analyzed (Participants) | 205 | 140
  ANTI-14, 6 months | 3.31 [2.92 to 3.75] | 0.06 [0.05 to 0.07]
  ANTI-14, 11-12 months: number analyzed (Participants) | 209 | 131
  ANTI-14, 11-12 months | 1.32 [1.13 to 1.54] | 0.04 [0.04 to 0.05]
  ANTI-14, 12-13 months: number analyzed (Participants) | 193 | 120
  ANTI-14, 12-13 months | 4.84 [4.26 to 5.51] | 0.06 [0.05 to 0.07]
  ANTI-14, 18-22 months: number analyzed (Participants) | 189 | 122
  ANTI-14, 18-22 months | 1.57 [1.32 to 1.86] | 0.12 [0.09 to 0.15]
  ANTI-18C, 6 months: number analyzed (Participants) | 205 | 141
  ANTI-18C, 6 months | 3.38 [2.88 to 3.95] | 0.04 [0.03 to 0.04]
  ANTI-18C, 11-12 months: number analyzed (Participants) | 209 | 132
  ANTI-18C, 11-12 months | 1.49 [1.29 to 1.73] | 0.03 [0.02 to 0.03]
  ANTI-18C, 12-13 months: number analyzed (Participants) | 193 | 124
  ANTI-18C, 12-13 months | 10.60 [9.48 to 11.84] | 0.03 [0.03 to 0.03]
  ANTI-18C, 18-22 months: number analyzed (Participants) | 189 | 120
  ANTI-18C, 18-22 months | 2.16 [1.89 to 2.48] | 0.04 [0.03 to 0.05]
  ANTI-19F, 6 months: number analyzed (Participants) | 205 | 140
  ANTI-19F, 6 months | 3.40 [2.92 to 3.97] | 0.06 [0.05 to 0.07]
  ANTI-19F, 11-12 months: number analyzed (Participants) | 209 | 133
  ANTI-19F, 11-12 months | 1.51 [1.29 to 1.75] | 0.03 [0.03 to 0.04]
  ANTI-19F, 12-13 months: number analyzed (Participants) | 193 | 124
  ANTI-19F, 12-13 months | 7.41 [6.54 to 8.40] | 0.04 [0.04 to 0.05]
  ANTI-19F, 18-22 months: number analyzed (Participants) | 189 | 123
  ANTI-19F, 18-22 months | 2.10 [1.79 to 2.47] | 0.07 [0.05 to 0.10]
  ANTI-23F, 6 months: number analyzed (Participants) | 205 | 142
  ANTI-23F, 6 months | 0.54 [0.45 to 0.65] | 0.04 [0.03 to 0.04]
  ANTI-23F, 11-12 months: number analyzed (Participants) | 209 | 134
  ANTI-23F, 11-12 months | 0.42 [0.35 to 0.50] | 0.03 [0.03 to 0.03]
  ANTI-23F, 12-13 months: number analyzed (Participants) | 193 | 123
  ANTI-23F, 12-13 months | 2.18 [1.88 to 2.54] | 0.03 [0.03 to 0.04]
  ANTI-23F, 18-22 months: number analyzed (Participants) | 189 | 122
  ANTI-23F, 18-22 months | 0.75 [0.63 to 0.88] | 0.04 [0.04 to 0.05]

64. Secondary Outcome: PNEUMOCOCCAL ANTIBODY CONCENTRATIONS AGAINST CROSS-REACTIVE PNEUMOCOCCAL SEROTYPES 6A AND 19A, IN THE IMMUNO SUBSET, IN SUBJECTS RECEIVING 3+1 INFANT SCHEDULES OF 10PN
Description: Antibody concentrations were measured by 22F-inhibitionenzyme-linked Immunosorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). Serotypes assessed were the cross-reactive pneumococcal serotypes 6A and 19A. The cut-off of the assay was >= 0.05 µg/mL. The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups.
Time Frame: as for outcome 62
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn3+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group
Number analyzed (Participants) | 208 | 122
µg/mL
  ANTI-6A, 6 months: number analyzed (Participants) | 208 | 120
  ANTI-6A, 6 months | 0.13 [0.11 to 0.15] | 0.03 [0.03 to 0.04]
  ANTI-6A, 11-12 months: number analyzed (Participants) | 202 | 121
  ANTI-6A, 11-12 months | 0.19 [0.16 to 0.23] | 0.03 [0.03 to 0.03]
  ANTI-6A, 12-13 months: number analyzed (Participants) | 189 | 120
  ANTI-6A, 12-13 months | 0.53 [0.43 to 0.65] | 0.03 [0.03 to 0.03]
  ANTI-6A, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-6A, 18-22 months | 0.30 [0.25 to 0.36] | 0.04 [0.03 to 0.05]
  ANTI-19A, 6 months: number analyzed (Participants) | 208 | 120
  ANTI-19A, 6 months | 0.15 [0.12 to 0.18] | 0.04 [0.04 to 0.05]
  ANTI-19A, 11-12 months: number analyzed (Participants) | 202 | 122
  ANTI-19A, 11-12 months | 0.23 [0.19 to 0.28] | 0.03 [0.03 to 0.03]
  ANTI-19A, 12-13 months: number analyzed (Participants) | 188 | 117
  ANTI-19A, 12-13 months | 0.95 [0.75 to 1.19] | 0.04 [0.03 to 0.05]
  ANTI-19A, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-19A, 18-22 months | 0.46 [0.38 to 0.55] | 0.06 [0.05 to 0.08]

65. Secondary Outcome: PNEUMOCOCCAL ANTIBODY CONCENTRATIONS AGAINST CROSS-REACTIVE PNEUMOCOCCAL SEROTYPES 6A AND 19A, IN THE IMMUNO SUBSET, IN SUBJECTS RECEIVING 2+1 INFANT SCHEDULES OF 10PN
Description: as for outcome 64
Time Frame: as for outcome 63
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn2+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group
Number analyzed (Participants) | 209 | 142
µg/mL
  ANTI-6A, 6 months: number analyzed (Participants) | 203 | 140
  ANTI-6A, 6 months | 0.09 [0.08 to 0.11] | 0.03 [0.03 to 0.04]
  ANTI-6A, 11-12 months: number analyzed (Participants) | 209 | 133
  ANTI-6A, 11-12 months | 0.14 [0.12 to 0.17] | 0.03 [0.03 to 0.03]
  ANTI-6A, 12-13 months: number analyzed (Participants) | 193 | 125
  ANTI-6A, 12-13 months | 0.50 [0.42 to 0.60] | 0.03 [0.03 to 0.04]
  ANTI-6A, 18-22 months: number analyzed (Participants) | 189 | 124
  ANTI-6A, 18-22 months | 0.27 [0.22 to 0.33] | 0.05 [0.04 to 0.06]
  ANTI-19A, 6 months: number analyzed (Participants) | 204 | 142
  ANTI-19A, 6 months | 0.13 [0.11 to 0.16] | 0.04 [0.04 to 0.05]
  ANTI-19A, 11-12 months: number analyzed (Participants) | 209 | 132
  ANTI-19A, 11-12 months | 0.15 [0.13 to 0.19] | 0.03 [0.03 to 0.03]
  ANTI-19A, 12-13 months: number analyzed (Participants) | 193 | 125
  ANTI-19A, 12-13 months | 0.89 [0.74 to 1.07] | 0.04 [0.03 to 0.04]
  ANTI-19A, 18-22 months: number analyzed (Participants) | 189 | 118
  ANTI-19A, 18-22 months | 0.36 [0.30 to 0.43] | 0.06 [0.05 to 0.08]

66. Secondary Outcome: TITERS FOR OPSONOPHAGOCYTIC ACTIVITY AGAINST VACCINE PNEUMOCOCCAL SEROTYPES, IN THE IMMUNO SUBSET, IN SUBJECTS RECEIVING 3+1 INFANT SCHEDULES OF 10PN
Description: Titers for opsonophagocytic activity against vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The cut-off of the assay was >= 8. The Immuno subset was constituted of the ± 1500 subjects from whom blood samples were collected, according to age and treatment groups.
Time Frame: as for outcome 62
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn3+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group
Number analyzed (Participants) | 202 | 120
Titers
  OPA-1, 6 months: number analyzed (Participants) | 202 | 118
  OPA-1, 6 months | 52.8 [40.7 to 68.4] | 4.1 [3.9 to 4.2]
  OPA-1, 11-12 months: number analyzed (Participants) | 199 | 119
  OPA-1, 11-12 months | 13.8 [10.8 to 17.6] | 4.4 [4.0 to 4.9]
  OPA-1, 12-13 months: number analyzed (Participants) | 184 | 120
  OPA-1, 12-13 months | 305.6 [238.9 to 390.8] | 4.6 [4.1 to 5.1]
  OPA-1, 18-22 months: number analyzed (Participants) | 184 | 112
  OPA-1, 18-22 months | 20.9 [16.1 to 27.1] | 4.1 [3.9 to 4.2]
  OPA-4, 6 months: number analyzed (Participants) | 199 | 112
  OPA-4, 6 months | 845.6 [746.8 to 957.4] | 4.6 [3.9 to 5.5]
  OPA-4, 11-12 months: number analyzed (Participants) | 190 | 119
  OPA-4, 11-12 months | 78.7 [61.1 to 101.3] | 6.0 [4.6 to 7.7]
  OPA-4, 12-13 months: number analyzed (Participants) | 184 | 115
  OPA-4, 12-13 months | 1745.7 [1476.3 to 2064.1] | 5.8 [4.5 to 7.5]
  OPA-4, 18-22 months: number analyzed (Participants) | 172 | 109
  OPA-4, 18-22 months | 105.1 [75.2 to 146.8] | 6.6 [4.9 to 8.8]
  OPA-5, 6 months: number analyzed (Participants) | 199 | 118
  OPA-5, 6 months | 65.9 [55.8 to 77.7] | 4.0 [4.0 to 4.1]
  OPA-5, 11-12 months: number analyzed (Participants) | 197 | 119
  OPA-5, 11-12 months | 20.6 [16.9 to 25.0] | 4.0 [4.0 to 4.0]
  OPA-5, 12-13 months: number analyzed (Participants) | 185 | 120
  OPA-5, 12-13 months | 191.6 [155.9 to 235.4] | 4.1 [3.9 to 4.2]
  OPA-5, 18-22 months: number analyzed (Participants) | 179 | 112
  OPA-5, 18-22 months | 26.9 [22.1 to 32.8] | 4.0 [4.0 to 4.0]
  OPA-6B, 6 months: number analyzed (Participants) | 195 | 111
  OPA-6B, 6 months | 740.6 [558.3 to 982.4] | 4.4 [3.8 to 5.0]
  OPA-6B, 11-12 months: number analyzed (Participants) | 181 | 116
  OPA-6B, 11-12 months | 220.3 [161.1 to 301.1] | 5.5 [4.2 to 7.2]
  OPA-6B, 12-13 months: number analyzed (Participants) | 181 | 117
  OPA-6B, 12-13 months | 736.3 [576.2 to 941.0] | 6.1 [4.6 to 8.2]
  OPA-6B, 18-22 months: number analyzed (Participants) | 179 | 106
  OPA-6B, 18-22 months | 75.0 [51.6 to 109.0] | 7.4 [5.3 to 10.4]
  OPA-7F, 6 months: number analyzed (Participants) | 197 | 103
  OPA-7F, 6 months | 3894.8 [3320.2 to 4569.0] | 87.6 [56.8 to 135.1]
  OPA-7F, 11-12 months: number analyzed (Participants) | 199 | 114
  OPA-7F, 11-12 months | 1960.7 [1654.4 to 2323.7] | 349.0 [252.2 to 483.0]
  OPA-7F, 12-13 months: number analyzed (Participants) | 184 | 117
  OPA-7F, 12-13 months | 5219.7 [4440.2 to 6136.0] | 436.7 [324.7 to 587.4]
  OPA-7F, 18-22 months: number analyzed (Participants) | 183 | 109
  OPA-7F, 18-22 months | 2124.5 [1813.8 to 2488.5] | 643.3 [479.5 to 863.0]
  OPA-9V, 6 months: number analyzed (Participants) | 194 | 112
  OPA-9V, 6 months | 2798.0 [2411.9 to 3246.0] | 6.5 [5.1 to 8.3]
  OPA-9V, 11-12 months: number analyzed (Participants) | 198 | 105
  OPA-9V, 11-12 months | 735.3 [625.6 to 864.3] | 19.4 [12.9 to 29.1]
  OPA-9V, 12-13 months: number analyzed (Participants) | 183 | 110
  OPA-9V, 12-13 months | 3491.2 [3049.2 to 3997.3] | 24.7 [16.0 to 38.0]
  OPA-9V, 18-22 months: number analyzed (Participants) | 181 | 100
  OPA-9V, 18-22 months | 809.1 [677.0 to 966.9] | 73.0 [44.9 to 118.5]
  OPA-14, 6 months: number analyzed (Participants) | 198 | 106
  OPA-14, 6 months | 1831.3 [1572.5 to 2132.7] | 10.5 [7.5 to 14.7]
  OPA-14, 11-12 months: number analyzed (Participants) | 198 | 105
  OPA-14, 11-12 months | 529.4 [446.6 to 627.6] | 18.9 [12.6 to 28.3]
  OPA-14, 12-13 months: number analyzed (Participants) | 185 | 109
  OPA-14, 12-13 months | 2657.2 [2280.6 to 3096.1] | 14.1 [9.3 to 21.3]
  OPA-14, 18-22 months: number analyzed (Participants) | 180 | 101
  OPA-14, 18-22 months | 639.0 [524.6 to 778.4] | 45.2 [27.4 to 74.4]
  OPA-18C, 6 months: number analyzed (Participants) | 192 | 116
  OPA-18C, 6 months | 543.3 [444.5 to 664.2] | 4.0 [4.0 to 4.0]
  OPA-18C, 11-12 months: number analyzed (Participants) | 195 | 118
  OPA-18C, 11-12 months | 50.0 [38.0 to 65.7] | 4.1 [3.9 to 4.3]
  OPA-18C, 12-13 months: number analyzed (Participants) | 183 | 118
  OPA-18C, 12-13 months | 1066.1 [890.3 to 1276.6] | 4.0 [4.0 to 4.0]
  OPA-18C, 18-22 months: number analyzed (Participants) | 179 | 110
  OPA-18C, 18-22 months | 70.4 [53.7 to 92.2] | 4.1 [3.9 to 4.4]
  OPA-19F, 6 months: number analyzed (Participants) | 196 | 118
  OPA-19F, 6 months | 649.6 [522.7 to 807.4] | 4.0 [4.0 to 4.0]
  OPA-19F, 11-12 months: number analyzed (Participants) | 198 | 117
  OPA-19F, 11-12 months | 63.5 [49.2 to 81.9] | 4.2 [3.9 to 4.6]
  OPA-19F, 12-13 months: number analyzed (Participants) | 183 | 119
  OPA-19F, 12-13 months | 1026.0 [807.3 to 1303.9] | 4.4 [3.9 to 4.8]
  OPA-19F, 18-22 months: number analyzed (Participants) | 181 | 110
  OPA-19F, 18-22 months | 80.1 [60.2 to 106.6] | 4.4 [4.0 to 4.8]
  OPA-23F, 6 months: number analyzed (Participants) | 196 | 111
  OPA-23F, 6 months | 1900.7 [1440.0 to 2508.7] | 7.0 [4.9 to 10.1]
  OPA-23F, 11-12 months: number analyzed (Participants) | 191 | 111
  OPA-23F, 11-12 months | 457.1 [313.4 to 666.8] | 15.9 [9.6 to 26.3]
  OPA-23F, 12-13 months: number analyzed (Participants) | 184 | 119
  OPA-23F, 12-13 months | 3248.2 [2705.9 to 3899.2] | 21.8 [12.9 to 37.0]
  OPA-23F, 18-22 months: number analyzed (Participants) | 174 | 109
  OPA-23F, 18-22 months | 398.6 [265.6 to 598.3] | 56.4 [29.9 to 106.3]

67. Secondary Outcome: TITERS FOR OPSONOPHAGOCYTIC ACTIVITY AGAINST VACCINE PNEUMOCOCCAL SEROTYPES, IN THE IMMUNO SUBSET, IN SUBJECTS RECEIVING 2+1 INFANT SCHEDULES OF 10PN
Description: Titers for opsonophagocytic activity against vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The cut-off of the assay was >= 8. The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups.
Time Frame: as for outcome 63
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn2+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group
Number analyzed (Participants) | 205 | 139
Titers
  OPA-1, 6 months: number analyzed (Participants) | 196 | 139
  OPA-1, 6 months | 38.3 [30.0 to 49.0] | 4.1 [3.9 to 4.2]
  OPA-1, 11-12 months: number analyzed (Participants) | 205 | 132
  OPA-1, 11-12 months | 9.8 [8.0 to 12.0] | 4.6 [4.0 to 5.3]
  OPA-1, 12-13 months: number analyzed (Participants) | 185 | 125
  OPA-1, 12-13 months | 256.9 [194.6 to 339.2] | 4.2 [3.9 to 4.5]
  OPA-1, 18-22 months: number analyzed (Participants) | 187 | 119
  OPA-1, 18-22 months | 13.0 [10.2 to 16.6] | 4.2 [4.0 to 4.5]
  OPA-4, 6 months: number analyzed (Participants) | 192 | 134
  OPA-4, 6 months | 553.0 [484.9 to 630.5] | 4.8 [4.1 to 5.6]
  OPA-4, 11-12 months: number analyzed (Participants) | 195 | 125
  OPA-4, 11-12 months | 43.4 [32.9 to 57.3] | 4.6 [4.0 to 5.2]
  OPA-4, 12-13 months: number analyzed (Participants) | 187 | 122
  OPA-4, 12-13 months | 1143.4 [961.9 to 1359.0] | 4.7 [4.0 to 5.6]
  OPA-4, 18-22 months: number analyzed (Participants) | 181 | 115
  OPA-4, 18-22 months | 51.9 [37.5 to 72.0] | 6.3 [5.0 to 7.9]
  OPA-5, 6 months: number analyzed (Participants) | 195 | 135
  OPA-5, 6 months | 48.5 [40.5 to 58.0] | 4.0 [4.0 to 4.0]
  OPA-5, 11-12 months: number analyzed (Participants) | 204 | 132
  OPA-5, 11-12 months | 15.6 [13.1 to 18.6] | 4.1 [3.9 to 4.3]
  OPA-5, 12-13 months: number analyzed (Participants) | 186 | 126
  OPA-5, 12-13 months | 145.6 [120.2 to 176.2] | 4.1 [3.9 to 4.3]
  OPA-5, 18-22 months: number analyzed (Participants) | 187 | 119
  OPA-5, 18-22 months | 21.2 [17.3 to 26.1] | 4.0 [4.0 to 4.0]
  OPA-6B, 6 months: number analyzed (Participants) | 186 | 132
  OPA-6B, 6 months | 268.6 [193.3 to 373.3] | 4.2 [3.8 to 4.7]
  OPA-6B, 11-12 months: number analyzed (Participants) | 191 | 130
  OPA-6B, 11-12 months | 121.6 [85.9 to 172.3] | 4.8 [4.0 to 5.9]
  OPA-6B, 12-13 months: number analyzed (Participants) | 183 | 117
  OPA-6B, 12-13 months | 879.1 [695.4 to 1111.2] | 5.3 [4.3 to 6.6]
  OPA-6B, 18-22 months: number analyzed (Participants) | 173 | 115
  OPA-6B, 18-22 months | 62.0 [41.6 to 92.3] | 7.9 [5.7 to 11.1]
  OPA-7F, 6 months: number analyzed (Participants) | 190 | 118
  OPA-7F, 6 months | 2553.5 [2124.7 to 3069.0] | 59.6 [38.3 to 92.6]
  OPA-7F, 11-12 months: number analyzed (Participants) | 202 | 124
  OPA-7F, 11-12 months | 1454.9 [1235.2 to 1713.7] | 364.8 [270.9 to 491.3]
  OPA-7F, 12-13 months: number analyzed (Participants) | 185 | 117
  OPA-7F, 12-13 months | 4863.2 [4211.1 to 5616.3] | 522.2 [372.4 to 732.3]
  OPA-7F, 18-22 months: number analyzed (Participants) | 186 | 113
  OPA-7F, 18-22 months | 2182.7 [1910.6 to 2493.5] | 856.5 [617.2 to 1188.6]
  OPA-9V, 6 months: number analyzed (Participants) | 186 | 130
  OPA-9V, 6 months | 1687.2 [1442.7 to 1973.1] | 5.3 [4.5 to 6.4]
  OPA-9V, 11-12 months: number analyzed (Participants) | 198 | 123
  OPA-9V, 11-12 months | 509.4 [431.3 to 601.6] | 19.3 [13.2 to 28.4]
  OPA-9V, 12-13 months: number analyzed (Participants) | 179 | 109
  OPA-9V, 12-13 months | 3196.0 [2718.4 to 3757.6] | 24.5 [15.9 to 37.6]
  OPA-9V, 18-22 months: number analyzed (Participants) | 185 | 108
  OPA-9V, 18-22 months | 700.1 [592.5 to 827.1] | 55.9 [35.4 to 88.2]
  OPA-14, 6 months: number analyzed (Participants) | 191 | 124
  OPA-14, 6 months | 1146.3 [944.2 to 1391.8] | 7.3 [5.5 to 9.5]
  OPA-14, 11-12 months: number analyzed (Participants) | 198 | 123
  OPA-14, 11-12 months | 233.5 [185.1 to 294.7] | 22.2 [14.8 to 33.1]
  OPA-14, 12-13 months: number analyzed (Participants) | 187 | 114
  OPA-14, 12-13 months | 1724.2 [1475.5 to 2014.8] | 26.2 [17.3 to 39.9]
  OPA-14, 18-22 months: number analyzed (Participants) | 182 | 104
  OPA-14, 18-22 months | 463.8 [380.9 to 564.7] | 99.2 [64.2 to 153.3]
  OPA-18C, 6 months: number analyzed (Participants) | 184 | 132
  OPA-18C, 6 months | 230.6 [177.0 to 300.4] | 4.0 [4.0 to 4.0]
  OPA-18C, 11-12 months: number analyzed (Participants) | 197 | 131
  OPA-18C, 11-12 months | 28.9 [21.6 to 38.6] | 4.1 [3.9 to 4.3]
  OPA-18C, 12-13 months: number analyzed (Participants) | 183 | 125
  OPA-18C, 12-13 months | 1052.2 [881.8 to 1255.5] | 4.2 [3.9 to 4.5]
  OPA-18C, 18-22 months: number analyzed (Participants) | 179 | 119
  OPA-18C, 18-22 months | 84.9 [63.4 to 113.6] | 6.2 [5.2 to 7.4]
  OPA-19F, 6 months: number analyzed (Participants) | 187 | 138
  OPA-19F, 6 months | 197.6 [148.6 to 262.8] | 4.1 [4.0 to 4.2]
  OPA-19F, 11-12 months: number analyzed (Participants) | 204 | 132
  OPA-19F, 11-12 months | 30.1 [23.6 to 38.5] | 4.2 [3.9 to 4.5]
  OPA-19F, 12-13 months: number analyzed (Participants) | 186 | 125
  OPA-19F, 12-13 months | 854.6 [672.1 to 1086.6] | 4.0 [4.0 to 4.0]
  OPA-19F, 18-22 months: number analyzed (Participants) | 187 | 116
  OPA-19F, 18-22 months | 56.7 [42.7 to 75.3] | 4.3 [4.0 to 4.7]
  OPA-23F, 6 months: number analyzed (Participants) | 188 | 131
  OPA-23F, 6 months | 897.1 [663.5 to 1212.9] | 5.6 [4.4 to 7.1]
  OPA-23F, 11-12 months: number analyzed (Participants) | 202 | 129
  OPA-23F, 11-12 months | 237.2 [156.6 to 359.3] | 17.3 [10.6 to 28.0]
  OPA-23F, 12-13 months: number analyzed (Participants) | 184 | 121
  OPA-23F, 12-13 months | 2630.7 [2047.9 to 3379.2] | 17.3 [10.6 to 28.2]
  OPA-23F, 18-22 months: number analyzed (Participants) | 181 | 113
  OPA-23F, 18-22 months | 222.7 [139.3 to 356.1] | 43.4 [23.8 to 79.0]

68. Secondary Outcome: TITERS FOR OPSONOPHAGOCYTIC ACTIVITY AGAINST CROSS-REACTIVE PNEUMOCOCCAL SEROTYPES 6A AND 19A, IN THE IMMUNO SUBSET. IN SUBJECTS RECEIVING 3+1 INFANT SCHEDULES OF 10PN
Description: Titers for opsonophagocytic activity against cross-reactive pneumococcal serotypes 6A and 19A. The cut-off of the assay was >= 8. The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups.
Time Frame: as for outcome 62
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn3+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group
Number analyzed (Participants) | 197 | 119
Titers
  OPA-6A, 6 months: number analyzed (Participants) | 191 | 116
  OPA-6A, 6 months | 90.8 [66.4 to 124.3] | 4.1 [3.9 to 4.4]
  OPA-6A, 11-12 months: number analyzed (Participants) | 188 | 117
  OPA-6A, 11-12 months | 70.9 [50.7 to 99.1] | 5.2 [4.2 to 6.4]
  OPA-6A, 12-13 months: number analyzed (Participants) | 177 | 115
  OPA-6A, 12-13 months | 173.8 [125.7 to 240.4] | 5.3 [4.3 to 6.5]
  OPA-6A, 18-22 months: number analyzed (Participants) | 179 | 109
  OPA-6A, 18-22 months | 32.9 [23.2 to 46.7] | 8.0 [5.9 to 11.0]
  OPA-19A, 6 months: number analyzed (Participants) | 193 | 118
  OPA-19A, 6 months | 25.2 [18.3 to 34.8] | 4.3 [3.9 to 4.8]
  OPA-19A, 11-12 months: number analyzed (Participants) | 197 | 118
  OPA-19A, 11-12 months | 8.6 [7.0 to 10.7] | 4.3 [3.9 to 4.8]
  OPA-19A, 12-13 months: number analyzed (Participants) | 181 | 119
  OPA-19A, 12-13 months | 145.0 [104.7 to 200.9] | 4.3 [4.0 to 4.8]
  OPA-19A, 18-22 months: number analyzed (Participants) | 182 | 111
  OPA-19A, 18-22 months | 12.2 [9.2 to 16.1] | 4.8 [4.1 to 5.7]

69. Secondary Outcome: TITERS FOR OPSONOPHAGOCYTIC ACTIVITY AGAINST CROSS-REACTIVE PNEUMOCOCCAL SEROTYPES 6A AND 19A, IN THE IMMUNO SUBSET. IN SUBJECTS RECEIVING 2+1 INFANT SCHEDULES OF 10PN
Description: as for outcome 68
Time Frame: as for outcome 63
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn2+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group
Number analyzed (Participants) | 204 | 137
Titers
  OPA-6A, 6 months: number analyzed (Participants) | 183 | 135
  OPA-6A, 6 months | 43.1 [31.2 to 59.5] | 4.4 [3.8 to 5.0]
  OPA-6A, 11-12 months: number analyzed (Participants) | 195 | 132
  OPA-6A, 11-12 months | 59.0 [42.0 to 82.9] | 5.1 [4.3 to 6.2]
  OPA-6A, 12-13 months: number analyzed (Participants) | 168 | 113
  OPA-6A, 12-13 months | 285.9 [205.3 to 398.2] | 5.3 [4.3 to 6.6]
  OPA-6A, 18-22 months: number analyzed (Participants) | 167 | 110
  OPA-6A, 18-22 months | 41.8 [28.8 to 60.8] | 10.5 [7.4 to 14.8]
  OPA-19A, 6 months: number analyzed (Participants) | 190 | 137
  OPA-19A, 6 months | 11.9 [9.2 to 15.5] | 4.1 [4.0 to 4.3]
  OPA-19A, 11-12 months: number analyzed (Participants) | 204 | 129
  OPA-19A, 11-12 months | 5.8 [5.0 to 6.9] | 4.0 [4.0 to 4.1]
  OPA-19A, 12-13 months: number analyzed (Participants) | 183 | 125
  OPA-19A, 12-13 months | 78.9 [55.5 to 112.2] | 4.1 [4.0 to 4.2]
  OPA-19A, 18-22 months: number analyzed (Participants) | 181 | 118
  OPA-19A, 18-22 months | 8.5 [6.6 to 10.9] | 5.1 [4.2 to 6.3]

70. Secondary Outcome: ANTIBODY CONCENTRATIONS AGAINST PROTEIN D (ANTI-PD), IN THE IMMUNO SUBSET. IN SUBJECTS RECEIVING 3+1 INFANT SCHEDULES OF 10PN
Description: ANTI-PD concentrations are expressed as geometric mean concentrations (GMCs), in enzyme-linked immunosorbent assay (ELISA) unit per milliliter (EL.U/mL). The cut-off of the assay was >= 100 EL.U/mL. The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups.
Time Frame: as for outcome 62
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10Pn3+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group
Number analyzed (Participants) | 209 | 123
EL.U/mL
  ANTI-PD, 6 months: number analyzed (Participants) | 209 | 121
  ANTI-PD, 6 months | 1869.4 [1670.7 to 2091.7] | 60.5 [54.8 to 66.7]
  ANTI-PD, 11-12 months: number analyzed (Participants) | 203 | 123
  ANTI-PD, 11-12 months | 955.2 [837.1 to 1089.9] | 62.7 [56.4 to 69.7]
  ANTI-PD, 12-13 months: number analyzed (Participants) | 188 | 118
  ANTI-PD, 12-13 months | 2734.7 [2406.0 to 3108.3] | 61.6 [55.0 to 69.0]
  ANTI-PD, 18-22 months: number analyzed (Participants) | 185 | 113
  ANTI-PD, 18-22 months | 1030.0 [884.3 to 1199.7] | 65.5 [57.4 to 74.8]

71. Secondary Outcome: ANTIBODY CONCENTRATIONS AGAINST PROTEIN D(ANTI-PD), IN THE IMMUNO SUBSET. IN SUBJECTS RECEIVING 2+1 INFANT SCHEDULES OF 10PN
Description: as for outcome 70
Time Frame: as for outcome 63
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10Pn2+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group
Number analyzed (Participants) | 209 | 139
EL.U/mL
  ANTI-PD, 6 months: number analyzed (Participants) | 203 | 139
  ANTI-PD, 6 months | 1062.9 [936.0 to 1207.0] | 66.1 [60.3 to 72.4]
  ANTI-PD, 11-12 months: number analyzed (Participants) | 209 | 131
  ANTI-PD, 11-12 months | 505.6 [439.2 to 582.1] | 62.9 [57.0 to 69.5]
  ANTI-PD, 12-13 months: number analyzed (Participants) | 193 | 127
  ANTI-PD, 12-13 months | 1903.9 [1642.7 to 2206.6] | 68.2 [61.1 to 76.1]
  ANTI-PD, 18-22 months: number analyzed (Participants) | 188 | 124
  ANTI-PD, 18-22 months | 687.7 [577.8 to 818.4] | 78.6 [68.8 to 89.8]

72. Secondary Outcome: PNEUMOCOCCAL ANTIBODY CONCENTRATIONS AGAINST PNEUMOCOCCAL VACCINE SEROTYPES, IN THE IMMUNO SUBSET. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: Antibody concentrations were measured by 22F-inhibitionenzyme-linked Immunosorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). Serotypes assessed were the pneumococcal vaccine serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The cut-off of the assay was >= 0.05 µg/mL. The Immuno subset was constituted of the first ± 1500 subjects from whom blood samples were collected, according to age and treatment groups.
Time Frame: At 8-12 months (mths) of age (1 mth post dose 1); at 9-13 mths of age (1 mth post dose 2) ; at 13-17 mths of age (pre-booster dose) ; at 14-18 mths of age ( 1 mths post-booster) ; at 23-27 mths of age (10 mths post-booster)
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 151 | 101
µg/mL
  ANTI-1, 9-13 months: number analyzed (Participants) | 151 | 100
  ANTI-1, 9-13 months | 1.96 [1.72 to 2.23] | 0.03 [0.03 to 0.03]
  ANTI-1, 13-17 months: number analyzed (Participants) | 144 | 97
  ANTI-1, 13-17 months | 0.66 [0.58 to 0.75] | 0.04 [0.03 to 0.05]
  ANTI-1, 14-18 months: number analyzed (Participants) | 137 | 90
  ANTI-1, 14-18 months | 2.62 [2.33 to 2.94] | 0.04 [0.03 to 0.05]
  ANTI-1, 23-27 months: number analyzed (Participants) | 124 | 88
  ANTI-1, 23-27 months | 0.59 [0.51 to 0.68] | 0.05 [0.04 to 0.06]
  ANTI-4, 9-13 months: number analyzed (Participants) | 150 | 101
  ANTI-4, 9-13 months | 5.85 [5.16 to 6.63] | 0.03 [0.02 to 0.03]
  ANTI-4, 13-17 months: number analyzed (Participants) | 144 | 96
  ANTI-4, 13-17 months | 1.55 [1.36 to 1.76] | 0.03 [0.02 to 0.03]
  ANTI-4, 14-18 months: number analyzed (Participants) | 135 | 90
  ANTI-4, 14-18 months | 5.45 [4.85 to 6.14] | 0.03 [0.02 to 0.03]
  ANTI-4, 23-27 months: number analyzed (Participants) | 124 | 88
  ANTI-4, 23-27 months | 1.21 [1.07 to 1.38] | 0.03 [0.03 to 0.03]
  ANTI-5, 9-13 months: number analyzed (Participants) | 151 | 99
  ANTI-5, 9-13 months | 2.40 [2.13 to 2.72] | 0.04 [0.03 to 0.04]
  ANTI-5, 13-17 months: number analyzed (Participants) | 144 | 96
  ANTI-5, 13-17 months | 1.19 [1.06 to 1.34] | 0.06 [0.05 to 0.07]
  ANTI-5, 14-18 months: number analyzed (Participants) | 137 | 89
  ANTI-5, 14-18 months | 4.11 [3.71 to 4.56] | 0.07 [0.05 to 0.08]
  ANTI-5, 23-27 months: number analyzed (Participants) | 123 | 87
  ANTI-5, 23-27 months | 1.30 [1.12 to 1.51] | 0.13 [0.09 to 0.17]
  ANTI-6B, 9-13 months: number analyzed (Participants) | 151 | 100
  ANTI-6B, 9-13 months | 0.27 [0.21 to 0.33] | 0.03 [0.03 to 0.03]
  ANTI-6B, 13-17 months: number analyzed (Participants) | 144 | 97
  ANTI-6B, 13-17 months | 0.49 [0.40 to 0.58] | 0.03 [0.03 to 0.04]
  ANTI-6B, 14-18 months: number analyzed (Participants) | 137 | 90
  ANTI-6B, 14-18 months | 1.06 [0.85 to 1.31] | 0.03 [0.03 to 0.04]
  ANTI-6B, 23-27 months: number analyzed (Participants) | 124 | 88
  ANTI-6B, 23-27 months | 0.52 [0.42 to 0.65] | 0.06 [0.04 to 0.07]
  ANTI-7F, 9-13 months: number analyzed (Participants) | 150 | 100
  ANTI-7F, 9-13 months | 3.61 [3.21 to 4.06] | 0.03 [0.03 to 0.03]
  ANTI-7F, 13-17 months: number analyzed (Participants) | 144 | 97
  ANTI-7F, 13-17 months | 2.22 [1.97 to 2.51] | 0.03 [0.03 to 0.04]
  ANTI-7F, 14-18 months: number analyzed (Participants) | 137 | 89
  ANTI-7F, 14-18 months | 5.44 [4.80 to 6.15] | 0.04 [0.03 to 0.05]
  ANTI-7F, 23-27 months: number analyzed (Participants) | 123 | 88
  ANTI-7F, 23-27 months | 2.08 [1.82 to 2.39] | 0.05 [0.04 to 0.06]
  ANTI-9V, 9-13 months: number analyzed (Participants) | 151 | 100
  ANTI-9V, 9-13 months | 1.42 [1.24 to 1.64] | 0.03 [0.02 to 0.03]
  ANTI-9V, 13-17 months: number analyzed (Participants) | 144 | 96
  ANTI-9V, 13-17 months | 0.88 [0.76 to 1.02] | 0.03 [0.03 to 0.04]
  ANTI-9V, 14-18 months: number analyzed (Participants) | 137 | 90
  ANTI-9V, 14-18 months | 2.81 [2.44 to 3.23] | 0.03 [0.03 to 0.04]
  ANTI-9V, 23-27 months: number analyzed (Participants) | 123 | 88
  ANTI-9V, 23-27 months | 1.16 [0.99 to 1.37] | 0.03 [0.03 to 0.04]
  ANTI-14, 9-13 months: number analyzed (Participants) | 150 | 100
  ANTI-14, 9-13 months | 3.81 [3.34 to 4.35] | 0.05 [0.04 to 0.06]
  ANTI-14, 13-17 months: number analyzed (Participants) | 144 | 95
  ANTI-14, 13-17 months | 3.06 [2.69 to 3.49] | 0.08 [0.06 to 0.11]
  ANTI-14, 14-18 months: number analyzed (Participants) | 137 | 89
  ANTI-14, 14-18 months | 8.38 [7.42 to 9.47] | 0.10 [0.07 to 0.14]
  ANTI-14, 23-27 months: number analyzed (Participants) | 123 | 88
  ANTI-14, 23-27 months | 2.91 [2.44 to 3.48] | 0.13 [0.09 to 0.19]
  ANTI-18C, 9-13 months: number analyzed (Participants) | 150 | 101
  ANTI-18C, 9-13 months | 10.03 [8.67 to 11.61] | 0.03 [0.03 to 0.03]
  ANTI-18C, 13-17 months: number analyzed (Participants) | 144 | 97
  ANTI-18C, 13-17 months | 4.70 [4.01 to 5.50] | 0.03 [0.03 to 0.04]
  ANTI-18C, 14-18 months: number analyzed (Participants) | 137 | 90
  ANTI-18C, 14-18 months | 19.87 [17.08 to 23.12] | 0.03 [0.03 to 0.04]
  ANTI-18C, 23-27 months: number analyzed (Participants) | 123 | 88
  ANTI-18C, 23-27 months | 5.46 [4.61 to 6.46] | 0.04 [0.03 to 0.06]
  ANTI-19F, 9-13 months: number analyzed (Participants) | 151 | 100
  ANTI-19F, 9-13 months | 6.64 [5.41 to 8.15] | 0.04 [0.03 to 0.05]
  ANTI-19F, 13-17 months: number analyzed (Participants) | 144 | 93
  ANTI-19F, 13-17 months | 3.41 [2.81 to 4.14] | 0.05 [0.04 to 0.07]
  ANTI-19F, 14-18 months: number analyzed (Participants) | 137 | 86
  ANTI-19F, 14-18 months | 11.73 [9.73 to 14.13] | 0.06 [0.04 to 0.08]
  ANTI-19F, 23-27 months: number analyzed (Participants) | 124 | 87
  ANTI-19F, 23-27 months | 3.69 [3.06 to 4.44] | 0.09 [0.07 to 0.13]
  ANTI-23F, 9-13 months: number analyzed (Participants) | 151 | 100
  ANTI-23F, 9-13 months | 0.55 [0.44 to 0.70] | 0.03 [0.03 to 0.03]
  ANTI-23F, 13-17 months: number analyzed (Participants) | 144 | 94
  ANTI-23F, 13-17 months | 0.64 [0.54 to 0.77] | 0.04 [0.03 to 0.05]
  ANTI-23F, 14-18 months: number analyzed (Participants) | 137 | 88
  ANTI-23F, 14-18 months | 2.04 [1.71 to 2.43] | 0.04 [0.03 to 0.05]
  ANTI-23F, 23-27 months: number analyzed (Participants) | 123 | 87
  ANTI-23F, 23-27 months | 0.80 [0.66 to 0.96] | 0.06 [0.05 to 0.08]

73. Secondary Outcome: PNEUMOCOCCAL ANTIBODY CONCENTRATIONS AGAINST PNEUMOCOCCAL VACCINE SEROTYPES, IN THE IMMUNO SUBSET. IN SUBJECTS RECEIVING RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 72
Time Frame: At 13-19 months (mths) of age (1 mth post dose 1); at 19-25 mths of age (1 mth post dose 2); at 21-27 mths of age (3 months post dose 2)
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 181 | 143
µg/mL
  ANTI-1, 13-19 months: number analyzed (Participants) | 181 | 138
  ANTI-1, 13-19 months | 0.73 [0.63 to 0.84] | 0.04 [0.04 to 0.05]
  ANTI-1, 19-25 months: number analyzed (Participants) | 167 | 134
  ANTI-1, 19-25 months | 1.87 [1.67 to 2.09] | 0.04 [0.03 to 0.04]
  ANTI-1, 21-27 months: number analyzed (Participants) | 162 | 132
  ANTI-1, 21-27 months | 0.95 [0.84 to 1.08] | 0.04 [0.04 to 0.05]
  ANTI-4, 13-19 months | 4.64 [4.11 to 5.25] | 0.03 [0.03 to 0.03]
  ANTI-4, 19-25 months: number analyzed (Participants) | 167 | 134
  ANTI-4, 19-25 months | 5.28 [4.77 to 5.84] | 0.03 [0.03 to 0.03]
  ANTI-4, 21-27 months: number analyzed (Participants) | 162 | 133
  ANTI-4, 21-27 months | 2.57 [2.29 to 2.87] | 0.03 [0.03 to 0.03]
  ANTI-5, 13-19 months: number analyzed (Participants) | 181 | 140
  ANTI-5, 13-19 months | 0.77 [0.67 to 0.88] | 0.07 [0.06 to 0.08]
  ANTI-5, 19-25 months: number analyzed (Participants) | 167 | 133
  ANTI-5, 19-25 months | 3.45 [3.05 to 3.90] | 0.07 [0.06 to 0.08]
  ANTI-5, 21-27 months: number analyzed (Participants) | 162 | 133
  ANTI-5, 21-27 months | 2.14 [1.88 to 2.44] | 0.08 [0.07 to 0.10]
  ANTI-6B, 13-19 months: number analyzed (Participants) | 181 | 136
  ANTI-6B, 13-19 months | 0.11 [0.09 to 0.13] | 0.04 [0.03 to 0.04]
  ANTI-6B, 19-25 months: number analyzed (Participants) | 167 | 133
  ANTI-6B, 19-25 months | 0.69 [0.57 to 0.83] | 0.05 [0.04 to 0.06]
  ANTI-6B, 21-27 months: number analyzed (Participants) | 162 | 133
  ANTI-6B, 21-27 months | 0.48 [0.40 to 0.57] | 0.06 [0.05 to 0.07]
  ANTI-7F, 13-19 months: number analyzed (Participants) | 181 | 142
  ANTI-7F, 13-19 months | 2.53 [2.22 to 2.89] | 0.03 [0.03 to 0.04]
  ANTI-7F, 19-25 months: number analyzed (Participants) | 167 | 134
  ANTI-7F, 19-25 months | 3.95 [3.58 to 4.35] | 0.04 [0.03 to 0.05]
  ANTI-7F, 21-27 months: number analyzed (Participants) | 162 | 133
  ANTI-7F, 21-27 months | 2.73 [2.48 to 3.01] | 0.05 [0.04 to 0.06]
  ANTI-9V, 13-19 months: number analyzed (Participants) | 181 | 140
  ANTI-9V, 13-19 months | 0.84 [0.73 to 0.97] | 0.03 [0.03 to 0.03]
  ANTI-9V, 19-25 months: number analyzed (Participants) | 167 | 134
  ANTI-9V, 19-25 months | 1.60 [1.42 to 1.81] | 0.03 [0.03 to 0.04]
  ANTI-9V, 21-27 months: number analyzed (Participants) | 163 | 129
  ANTI-9V, 21-27 months | 1.22 [1.07 to 1.39] | 0.03 [0.03 to 0.04]
  ANTI-14, 13-19 months | 1.07 [0.90 to 1.28] | 0.06 [0.05 to 0.08]
  ANTI-14, 19-25 months: number analyzed (Participants) | 167 | 132
  ANTI-14, 19-25 months | 6.04 [5.37 to 6.79] | 0.09 [0.07 to 0.12]
  ANTI-14, 21-27 months: number analyzed (Participants) | 161 | 133
  ANTI-14, 21-27 months | 3.73 [3.30 to 4.21] | 0.21 [0.15 to 0.29]
  ANTI-18C, 13-19 months: number analyzed (Participants) | 181 | 142
  ANTI-18C, 13-19 months | 3.76 [3.35 to 4.22] | 0.04 [0.03 to 0.04]
  ANTI-18C, 19-25 months: number analyzed (Participants) | 166 | 134
  ANTI-18C, 19-25 months | 21.27 [18.70 to 24.19] | 0.04 [0.03 to 0.04]
  ANTI-18C, 21-27 months: number analyzed (Participants) | 162 | 133
  ANTI-18C, 21-27 months | 12.44 [10.88 to 14.22] | 0.04 [0.03 to 0.05]
  ANTI-19F, 13-19 months | 2.63 [2.24 to 3.10] | 0.06 [0.05 to 0.08]
  ANTI-19F, 19-25 months: number analyzed (Participants) | 166 | 134
  ANTI-19F, 19-25 months | 12.10 [10.38 to 14.11] | 0.09 [0.07 to 0.12]
  ANTI-19F, 21-27 months: number analyzed (Participants) | 162 | 132
  ANTI-19F, 21-27 months | 8.49 [7.39 to 9.74] | 0.11 [0.08 to 0.15]
  ANTI-23F, 13-19 months: number analyzed (Participants) | 181 | 138
  ANTI-23F, 13-19 months | 0.16 [0.13 to 0.19] | 0.03 [0.03 to 0.04]
  ANTI-23F, 19-25 months: number analyzed (Participants) | 167 | 134
  ANTI-23F, 19-25 months | 1.27 [1.07 to 1.50] | 0.05 [0.04 to 0.06]
  ANTI-23F, 21-27 months: number analyzed (Participants) | 162 | 132
  ANTI-23F, 21-27 months | 0.83 [0.70 to 0.99] | 0.05 [0.04 to 0.06]

74. Secondary Outcome: PNEUMOCOCCAL ANTIBODY CONCENTRATIONS AGAINST CROSS-REACTIVE PNEUMOCOCCAL SEROTYPES, IN THE IMMUNO SUBSET. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 64
Time Frame: as for outcome 72
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 151 | 100
µg/mL
  ANTI-6A, 9-13 months: number analyzed (Participants) | 150 | 99
  ANTI-6A, 9-13 months | 0.11 [0.09 to 0.14] | 0.03 [0.03 to 0.03]
  ANTI-6A, 13-17 months: number analyzed (Participants) | 144 | 96
  ANTI-6A, 13-17 months | 0.23 [0.18 to 0.29] | 0.03 [0.03 to 0.04]
  ANTI-6A, 14.18 months: number analyzed (Participants) | 137 | 89
  ANTI-6A, 14.18 months | 0.70 [0.55 to 0.90] | 0.03 [0.03 to 0.04]
  ANTI-6A, 23-27 months: number analyzed (Participants) | 123 | 88
  ANTI-6A, 23-27 months | 0.33 [0.26 to 0.41] | 0.06 [0.04 to 0.07]
  ANTI-19A, 9-13 months | 0.33 [0.26 to 0.42] | 0.04 [0.03 to 0.04]
  ANTI-19A, 13-17 months: number analyzed (Participants) | 144 | 97
  ANTI-19A, 13-17 months | 0.49 [0.39 to 0.62] | 0.05 [0.04 to 0.06]
  ANTI-19A, 14.18 months: number analyzed (Participants) | 137 | 90
  ANTI-19A, 14.18 months | 1.98 [1.53 to 2.56] | 0.04 [0.04 to 0.06]
  ANTI-19A, 23-27 months: number analyzed (Participants) | 123 | 88
  ANTI-19A, 23-27 months | 0.93 [0.70 to 1.23] | 0.08 [0.06 to 0.11]

75. Secondary Outcome: PNEUMOCOCCAL ANTIBODY CONCENTRATIONS AGAINST CROSS-REACTIVE PNEUMOCOCCAL SEROTYPES, IN THE IMMUNO SUBSET. IN SUBJECTS RECEIVING RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 64
Time Frame: as for outcome 73
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 181 | 143
µg/mL
  ANTI-6A, 13-19 months | 0.06 [0.05 to 0.08] | 0.04 [0.03 to 0.04]
  ANTI-6A, 19-25 months: number analyzed (Participants) | 167 | 134
  ANTI-6A, 19-25 months | 0.32 [0.26 to 0.41] | 0.05 [0.04 to 0.06]
  ANTI-6A, 21-27 months: number analyzed (Participants) | 162 | 132
  ANTI-6A, 21-27 months | 0.29 [0.23 to 0.36] | 0.06 [0.05 to 0.08]
  ANTI-19A, 13-19 months: number analyzed (Participants) | 181 | 136
  ANTI-19A, 13-19 months | 0.20 [0.16 to 0.25] | 0.05 [0.04 to 0.06]
  ANTI-19A, 19-25 months: number analyzed (Participants) | 167 | 134
  ANTI-19A, 19-25 months | 2.61 [2.12 to 3.22] | 0.06 [0.05 to 0.07]
  ANTI-19A, 21-27 months: number analyzed (Participants) | 162 | 132
  ANTI-19A, 21-27 months | 1.72 [1.41 to 2.10] | 0.07 [0.05 to 0.09]

76. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH ACUTE OTITIS MEDIA (AOM) EPISODE ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: The PYAR (Person-Year Rate) as regards subjects with AOM episode was tabulated. PYAR was calculated as follows n (= number of subjects reported with event) divided by T (= sum of follow-up period expressed in years) (per 1000). An AOM episode assessed as with level 1 of diagnostic certainty was defined as an AOM event diagnosed by a physician according to the Finnish AOM management guidelines (confirmed cases) and reported by subjects' parent(s)/guardian(s) regardless the documentation in medical records or other source document. Note that a post-hoc re-analysis of AOM endpoints with a corrected definition of follow-up taking into account individual end of follow-up time was performed; the results of re-analysis as the most prominent for AOM outcome are presented in this summary.
Time Frame: Period of follow-up was anytime after the administration of first vaccine dose till the end of the blinded invasive disease (ID) follow-up period (31 January 2012).
Population: The total vaccinated cohort for analysis of AOM/RTI effectiveness included all vaccinated subjects for whom data concerning AOM/RTI effectiveness outcome measures were available.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1846 | 942 | 1329
Participants per 1000 person-years | 420.645 [396.814 to 445.534] | 415.560 [382.673 to 450.518] | 443.411 [414.786 to 473.491]

77. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH ACUTE OTITIS MEDIA (AOM) EPISODE ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 76
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 191 | 96
Participants per 1000 person-years | 510.388 [422.105 to 611.686] | 590.118 [460.887 to 744.354]

78. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH ACUTE OTITIS MEDIA (AOM) EPISODE ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 76
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 286 | 106
Participants per 1000 person-years | 598.065 [502.777 to 706.159] | 567.194 [419.613 to 749.861]

79. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH RECURRENT ACUTE OTITIS MEDIA (AOM) EPISODES ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: as for outcome 76
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1846 | 942 | 1329
Participants per 1000 person-years | 100.550 [89.076 to 113.091] | 103.008 [86.977 to 121.137] | 94.946 [81.957 to 109.407]

80. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH RECURRENT ACUTE OTITIS MEDIA (AOM) EPISODES ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 76
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 191 | 96
Participants per 1000 person-years | 78.521 [46.537 to 124.097] | 132.984 [76.012 to 215.958]

81. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH RECURRENT ACUTE OTITIS MEDIA (AOM) EPISODES ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 76
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 286 | 106
Participants per 1000 person-years | 90.355 [55.931 to 138.117] | 46.302 [12.616 to 118.550]

82. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH ACUTE OTITIS MEDIA (AOM) EPISODE ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY AND ACCOMPANIED WITH DOCUMENTED ANTIMICROBIAL PRESCRIPTION. IN SUBJECTS RECEIVING 3+1 AND 2+1 INFANT SCHEDULES OF 10PN
Description: as for outcome 76
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl-6W-6M/053 Group
Number analyzed (Participants) | 1846 | 942 | 1329
Participants per 1000 person-years | 409.795 [386.277 to 434.369] | 408.505 [375.904 to 443.176] | 430.984 [402.769 to 460.653]

83. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH ACUTE OTITIS MEDIA (AOM) EPISODE ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY AND ACCOMPANIED WITH DOCUMENTED ANTIMICROBIAL PRESCRIPTION. IN SUBJECTS RECEIVING 7-11M SCHEDULE OF 10PN
Description: as for outcome 76
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group
Number analyzed (Participants) | 191 | 96
Participants per 1000 person-years | 497.301 [410.212 to 597.410] | 581.807 [453.547 to 735.078]

84. Secondary Outcome: PERSON YEAR RATE AS REGARDS SUBJECTS WITH ACUTE OTITIS MEDIA (AOM) EPISODE ASSESSED AS WITH LEVEL 1 OF DIAGNOSTIC CERTAINTY AND ACCOMPANIED WITH DOCUMENTED ANTIMICROBIAL PRESCRIPTION. IN SUBJECTS RECEIVING 12-18M SCHEDULE OF 10PN
Description: as for outcome 76
Time Frame: as for outcome 76
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
Number analyzed (Participants) | 286 | 106
Participants per 1000 person-years | 593.763 [498.833 to 701.499] | 555.619 [409.670 to 736.670]

85. Secondary Outcome: Culture-confirmed Invasive Disease (ID) Person Year Rate - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course Till End of LT FU Period.
Description: as for outcome 3
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end of the long-term Follow-up period (The Follow-up period lasted at least 77 months).
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10272 | 10201
Participants per 1000 person-years
  Culture confirmed ID | 0.046 [0.013 to 0.118] | 0.268 [0.170 to 0.402]
  Pneumococcal invasive disease (IPD) | 0.023 [0.003 to 0.084] | 0.210 [0.124 to 0.331]
  Vaccine serotypes (vaccine type-IPD) | 0.0 [0.0 to 0.043] | 0.140 [0.072 to 0.244]
  Serotype 4 | 0.0 [0.0 to 0.043] | 0.0 [0.0 to 0.043]
  Serotype 6B | 0.0 [0.0 to 0.043] | 0.058 [0.019 to 0.136]
  Serotype 7F | 0.0 [0.0 to 0.043] | 0.0 [0.0 to 0.043]
  Serotype 14 | 0.0 [0.0 to 0.043] | 0.047 [0.013 to 0.119]
  Serotype 18C | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Serotype 19F | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Serotype 23F | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Cross-reactive serotypes | 0.012 [0.0 to 0.064] | 0.047 [0.013 to 0.119]
  Serotype 6A | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Serotype 19A | 0.012 [0.0 to 0.064] | 0.035 [0.007 to 0.102]
  Other pneumococcal serotypes | 0.012 [0.0 to 0.064] | 0.023 [0.003 to 0.084]
  Serotype 3 | 0.012 [0.0 to 0.064] | 0.012 [0.0 to 0.065]
  Serotype 12F | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Serotype 15C | 0.0 [0.0 to 0.043] | 0.0 [0.0 to 0.043]
  H. influenzae ID | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Non-typeable (NTHI) | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Other bacteria | 0.023 [0.003 to 0.084] | 0.058 [0.019 to 0.136]
  Neisseria meningitidis | 0.023 [0.003 to 0.084] | 0.023 [0.003 to 0.084]
  Streptococcus pyogenes | 0.0 [0.0 to 0.043] | 0.023 [0.003 to 0.084]
  Moraxella catarrhalis | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]

86. Secondary Outcome: Culture-confirmed Invasive Disease (ID) Person Year Rate - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course Till End of LT FU Period.
Description: as for outcome 3
Time Frame: as for outcome 85
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10053 | 10201
Participants per 1000 person-years
  Culture confirmed ID | 0.047 [0.013 to 0.122] | 0.268 [0.170 to 0.402]
  Pneumococcal invasive disease (IPD) | 0.024 [0.003 to 0.086] | 0.210 [0.124 to 0.331]
  Vaccine serotypes (vaccine type-IPD) | 0.012 [0.0 to 0.066] | 0.140 [0.072 to 0.244]
  Serotype 4 | 0.0 [0.0 to 0.044] | 0.0 [0.0 to 0.043]
  Serotype 6B | 0.0 [0.0 to 0.044] | 0.058 [0.019 to 0.136]
  Serotype 7F | 0.012 [0.0 to 0.066] | 0.0 [0.0 to 0.043]
  Serotype 14 | 0.0 [0.0 to 0.044] | 0.047 [0.013 to 0.119]
  Serotype 18C | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Serotype 19F | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Serotype 23F | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Cross-reactive serotypes | 0.0 [0.0 to 0.044] | 0.047 [0.013 to 0.119]
  Serotype 6A | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Serotype 19A | 0.0 [0.0 to 0.044] | 0.035 [0.007 to 0.102]
  Other pneumococcal serotypes | 0.012 [0.0 to 0.066] | 0.023 [0.003 to 0.084]
  Serotype 3 | 0.012 [0.0 to 0.066] | 0.012 [0.0 to 0.065]
  Serotype 12F | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Serotype 15C | 0.0 [0.0 to 0.044] | 0.0 [0.0 to 0.043]
  H. influenzae ID | 0.012 [0.0 to 0.066] | 0.012 [0.0 to 0.065]
  Non-typeable (NTHI) | 0.012 [0.0 to 0.066] | 0.012 [0.0 to 0.065]
  Other bacteria | 0.012 [0.0 to 0.066] | 0.058 [0.019 to 0.136]
  Neisseria meningitidis | 0.012 [0.0 to 0.066] | 0.023 [0.003 to 0.084]
  Streptococcus pyogenes | 0.0 [0.0 to 0.044] | 0.023 [0.003 to 0.084]
  Moraxella catarrhalis | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs: 4-day (Days 0-3) and 31-day (Days 0-30) post primary (PRI)/booster (BST) vaccination dose(s); SAEs: from day to study end, Month (M) 18 for 6W-6M groups, M16 for 7-11M groups and M9 for M12-18 groups.
Description: To avoid inconsistency between the AE reporting and the acute otitis media (AOM) questionnaire filled in by subjects' parent(s)/LAR(s), otitis was not reported as an AE if already reported via the AOM questionnaire.
Arm/Group | 10Pn3+1-6W-6M/053 Group | 10Pn2+1-6W-6M/053 Group | Ctrl3+1-6W-6M/053 Group | Ctrl2+1-6W-6M/053 Group | 10Pn7-11M/053 Group | Ctrl7-11M/053 Group | 10Pn12-18M/053 Group | Ctrl12-18M/053 Group
All-Cause Mortality (participants affected / at risk) | 0/1849 | 1/1316 | 0/1069 | 0/859 | 0/241 | 0/204 | 0/368 | 0/271
Serious Adverse Events (participants affected / at risk) | 163/1849 | 96/1316 | 77/1069 | 74/859 | 24/241 | 18/204 | 23/368 | 14/271
Other Adverse Events (participants affected / at risk) | 1840/1849 | 1295/1316 | 1038/1069 | 805/859 | 232/241 | 193/204 | 354/368 | 254/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10Pn3+1-6W-6M/053 Group (N=1849) | 10Pn2+1-6W-6M/053 Group (N=1316) | Ctrl3+1-6W-6M/053 Group (N=1069) | Ctrl2+1-6W-6M/053 Group (N=859) | 10Pn7-11M/053 Group (N=241) | Ctrl7-11M/053 Group (N=204) | 10Pn12-18M/053 Group (N=368) | Ctrl12-18M/053 Group (N=271)
Bronchitis (Infections and infestations) | 33 | 13 | 19 | 20 | 9 | 5 | 5 | 2
Otitis media (Infections and infestations) | 22 | 7 | 9 | 13 | 1 | 0 | 1 | 2
Bronchiolitis (Infections and infestations) | 9 | 8 | 5 | 9 | 1 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 15 | 7 | 5 | 4 | 3 | 1 | 2 | 1
Laryngitis (Infections and infestations) | 12 | 6 | 4 | 7 | 1 | 0 | 2 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 11 | 7 | 4 | 4 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 10 | 5 | 3 | 5 | 1 | 1 | 2 | 1
Pyelonephritis (Infections and infestations) | 10 | 7 | 2 | 2 | 0 | 1 | 2 | 1
Febrile convulsion (Nervous system disorders) | 5 | 6 | 1 | 2 | 0 | 1 | 2 | 1
Pyrexia (General disorders) | 4 | 4 | 4 | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 3 | 3 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4 | 3 | 4 | 1 | 4 | 2
Otitis media acute (Infections and infestations) | 5 | 2 | 1 | 3 | 2 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 5 | 2 | 2 | 1 | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0
Infection (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Adenovirus infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Amaurotic familial idiocy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 7 | 2 | 4 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Combined immunodeficiency (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Craniosynostosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis adenovirus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperreflexia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngomalcia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 3 | 4 | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 4 | 0 | 1 | 3 | 0 | 2 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 2 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Crying (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Developmental delay (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Krabbe's disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mitochondrial encephalomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Septic arthritis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Roseola (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Accidental drug intake by child (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis orbital (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.98% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10Pn3+1-6W-6M/053 Group (N=1849) | 10Pn2+1-6W-6M/053 Group (N=1316) | Ctrl3+1-6W-6M/053 Group (N=1069) | Ctrl2+1-6W-6M/053 Group (N=859) | 10Pn7-11M/053 Group (N=241) | Ctrl7-11M/053 Group (N=204) | 10Pn12-18M/053 Group (N=368) | Ctrl12-18M/053 Group (N=271)
Diarrhoea (Gastrointestinal disorders) | 140 (160) | 78 (86) | 75 (84) | 52 (58) | 22 (27) | 17 (19) | 26 (28) | 25 (28)
Teething (Gastrointestinal disorders) | 66 (83) | 40 (45) | 61 (70) | 34 (39) | 11 (15) | 21 (21) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 419 (720) | 239 (340) | 71 (89) | 29 (34) | 30 (47) | 5 (6) | 45 (52) | 2 (2)
Pain (General disorders) | 1399 (2898) | 983 (1830) | 396 (614) | 275 (374) | 176 (351) | 76 (111) | 301 (463) | 116 (143)
Pyrexia (General disorders) | 1030 (1621) | 688 (1062) | 377 (483) | 261 (334) | 115 (154) | 68 (77) | 119 (143) | 62 (70)
Swelling (General disorders) | 1257 (2716) | 878 (1594) | 382 (575) | 205 (262) | 154 (290) | 50 (68) | 209 (290) | 42 (51)
Nasopharyngitis (Infections and infestations) | 107 (127) | 49 (59) | 64 (87) | 64 (74) | 18 (19) | 11 (14) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 69 (80) | 32 (34) | 57 (65) | 24 (24) | 25 (26) | 19 (23) | 25 (29) | 22 (23)
Rhinitis (Infections and infestations) | 147 (178) | 74 (88) | 105 (123) | 72 (83) | 21 (25) | 36 (43) | 29 (33) | 25 (29)
Upper respiratory tract infection (Infections and infestations) | 233 (291) | 109 (122) | 131 (161) | 45 (53) | 38 (46) | 50 (67) | 36 (37) | 40 (47)
Decreased appetite (Metabolism and nutrition disorders) | 1103 (1832) | 713 (1072) | 527 (828) | 356 (483) | 153 (217) | 105 (159) | 191 (238) | 118 (140)
Somnolence (Nervous system disorders) | 1493 (3305) | 1024 (1876) | 723 (1394) | 539 (887) | 165 (286) | 101 (161) | 214 (281) | 118 (145)
Irritability (Psychiatric disorders) | 1761 (4864) | 1204 (2592) | 914 (2134) | 688 (1304) | 207 (428) | 152 (272) | 283 (407) | 142 (181)
Erythema (Skin and subcutaneous tissue disorders) | 1522 (3821) | 1042 (2077) | 584 (1188) | 397 (665) | 182 (369) | 89 (162) | 265 (398) | 130 (179)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 7 (7) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 12 (13) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 11 (13) | 14 (16) | 15 (16)

LIMITATIONS AND CAVEATS:
Number allocation errors were identified for 3 subjects after Dose 1, which GSK assessed as not having significant impact. Lower & upper respiratory tract infections endpoint results are not presented, being uninterpretable due to low sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.